CLINICAL TRIAL: NCT03919799
Title: A Phase 2, Randomized, Placebo-controlled, Double-blind, Open-label Extension Multicenter Study to Evaluate the Efficacy and Safety of Belumosudil (KD025) in Subjects With Diffuse Cutaneous Systemic Sclerosis
Brief Title: KD025 in Subjects With Diffuse Cutaneous Systemic Sclerosis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision due to slow enrollment and strategic consideration; not driven by any safety concerns.
Sponsor: Kadmon, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC17665; KD025-209 (Other: Kadmon)
Record Dates: First submitted 2018-11-21; First posted 2019-04-18 (Actual); Results first posted 2023-08-30 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: System; Sclerosis; Diffuse Cutaneous Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Diffuse | interventions — belumosudil; KD025

STUDY DESIGN:
Intervention Model Description: Three groups (1:1:1) to receive orally administered belumosudil 200 mg QD, belumosudil 200 mg BID, or matched placebo for 28 weeks. The study was double-blinded for the first 28 weeks followed by an open-label extension of 24 weeks.
  After unblinding, the participants in the belumosudil groups continued on the same belumosudil dose whereas the participants in the placebo group were re-randomized to one of the belumosudil doses (200 mg QD or 200 BID) in 1:1 fashion.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blinded for the first 28 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Belumosudil QD/Belumosudil QD (Experimental): Participants received belumosudil 200 mg tablet, QD orally for 28 weeks during the DB period. After completion of DB period, participants entered open-label extension (OLE) period and continued to receive belumosudil 200 mg tablet QD orally for 24 weeks in OLE period (i.e., up to Week 52).
  Interventions: Drug: Belumosudil (KD025)
- Belumosudil BID/Belumosudil BID (Experimental): Participants received belumosudil 200 mg tablet BID orally, for 28 weeks during the DB period. After completion of DB period, participants entered OLE period and continued to receive belumosudil 200 mg tablet BID orally for 24 weeks in OLE period (i.e., up to Week 52).
  Interventions: Drug: Belumosudil (KD025)
- DB Period: Placebo (Placebo Comparator): Participants received placebo (matched to belumosudil) tablet, orally for 28 weeks during the DB period.
  Interventions: Drug: Placebo
- OLE Period: Placebo/Belumosudil QD (Experimental): Participants who had received placebo in the DB period were entered and re-randomized into OLE period and received belumosudil 200 mg tablet QD orally for 24 weeks (i.e., up to Week 52) in the OLE period.
  Interventions: Drug: Belumosudil (KD025)
- OLE Period: Placebo/Belumosudil BID (Experimental): Participants who had received placebo in the DB period were entered and re-randomized into OLE period and received belumosudil 200 mg tablet BID orally for 24 weeks (i.e., up to Week 52) in the OLE period.
  Interventions: Drug: Belumosudil (KD025)

INTERVENTIONS:
Drug: Belumosudil (KD025) — ROCK-2 Inhibitor
  Arms: Belumosudil BID/Belumosudil BID; Belumosudil QD/Belumosudil QD; OLE Period: Placebo/Belumosudil BID; OLE Period: Placebo/Belumosudil QD
Drug: Placebo — Inactive substance
  Arms: DB Period: Placebo

SUMMARY:
This randomized, placebo-controlled phase 2 study was seeking to evaluate the efficacy and safety of belumosudil (KD025) for the treatment of diffuse cutaneous systematic sclerosis. Enrolment was terminated earlier than planned for business reasons unrelated to safety. A total of 36 participants were enrolled and randomized into 3 groups to either receive orally administered belumosudil (200 milligrams [mg] once daily [QD] and 200 mg twice daily [BID]) or matched placebo in 1:1:1 ratio in the double-blind (DB) period of this study. Study drug dosing was for 52 weeks: double-blinded for the first 28 weeks followed by an open-label extension of 24 weeks. After unblinding, the participants on belumosudil continued on the same belumosudil dose whereas the participants in the placebo group were re-randomized to one of the belumosudil doses in a 1:1 ratio.

DETAILED DESCRIPTION:
Systemic sclerosis (SSc) is a chronic autoimmune disease that causes widespread microvascular damage and excessive deposition of collagen in the skin and internal organs. Limited cutaneous systemic sclerosis is primarily cutaneous, affecting the hands, arms, and face. Diffuse cutaneous systemic sclerosis (dcSSc) is a more serious manifestation of the disease and is often rapidly progressive, not only involving the skin, but also involving internal organs including kidney, heart, and lungs.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants greater than or equal to (>=) 18 years old with the diagnosis of dcSSc according to the 2013 American College of Rheumatology and European League Against Rheumatism criteria.
2. Had disease duration (defined as interval from first non-Raynaud disease manifestation) of less than or equal to (<=) 5 years.
3. Had mRSS of >= 15 but <= 35.
4. Active disease defined as any of the following within the 6 months prior to screening:

   1. Increase in mRSS by >= 3 units.
   2. Increase in mRSS by >= 2 units with involvement of 1 new body area.
   3. Involvement of 2 new body areas.
   4. Symptoms indicative of skin activity such as severe cutaneous itching or burning.
5. Participants who had received concomitant immunosuppression must be on a stable dose for at least 3 months prior to screening.
6. Adequate organ and bone marrow functions evaluated during the 28 days prior to enrollment as follows:

   1. Absolute neutrophil count >= 1.5*10^9/L.
   2. Platelet count >=100*10^9/L.
   3. Total bilirubin <= 1.0*upper limit of normal (ULN).
   4. Alanine aminotransferase (ALT), aspartate aminotransferase (AST), and serum creatinine <= 1.5*ULN.
7. Female participants of childbearing potential had a negative pregnancy test at screening. Females of childbearing potential were defined as sexually mature women without prior hysterectomy or who have had any evidence of menses in the past 12 months. However, women who had been amenorrheic for 12 or more months were still considered to be of childbearing potential if the amenorrhea was possibly due to prior chemotherapy, anti-estrogens, or ovarian suppression.

   1. Women of childbearing potential (i.e., menstruating women) had a negative urine pregnancy test (positive urine tests were to be confirmed by serum test) documented within the 24-hour period prior to the first dose of study drug.
   2. Sexually active women of childbearing potential enrolled in the study must agree to use 2 forms of accepted methods of contraception during the course of the study and for 3 months after their last dose of study drug. Effective birth control includes (1) intrauterine device plus 1 barrier method; (2) on stable doses of hormonal contraception for at least 3 months (e.g., oral, injectable, implant, transdermal) plus 1 barrier method; or (3) two barrier methods. Effective barrier methods were male or female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm), or a vasectomized partner.
8. For male participants who were sexually active and who were partners of premenopausal women, agreement to use 2 forms of contraception as in Criterion Number 7 above during the treatment period and for at least 3 months after the last dose of study drug.
9. Male participants must not donate sperm for 3 months after last dose of study drug.
10. Able to provide written informed consent prior to the performance of any study-specific procedures.

Exclusion Criteria:

1. Participant had corrected QT interval QTcF greater than (>) 450 milliseconds.
2. Ongoing use or current use of concomitant medication known to have the potential for QTc prolongation.
3. Female participant who was pregnant or breastfeeding.
4. Participated in another study with an investigational drug within 28 days of study entry (for studies involving biologics within 3 half-lives of the biologic).
5. History or other evidence of severe illness or any other conditions that would make the participant, in the opinion of the Investigator, unsuitable for the study.
6. Chronic heart failure with New York Heart Association Class II, III, or IV.
7. Acute or chronic liver disease (e.g., cirrhosis).
8. Positive human immunodeficiency virus (HIV) test.
9. Active hepatitis C virus (HCV), hepatitis B virus (HBV), or positive whole blood tuberculin test.
10. Diagnosed with any malignancy within 3 years of enrollment, with the exception of basal cell or completely resected squamous cell carcinoma of the skin, resected in situ cervical malignancy, resected breast ductal carcinoma in situ, or low-risk prostate cancer after curative resection.
11. Has had previous exposure to belumosudil or known allergy/sensitivity to belumosudil, or any other ROCK2 inhibitor.
12. Scleroderma renal crisis within 4 months prior to enrollment.
13. FVC <= 50% Predicted.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2022-08-09 (Actual); Study Completion 2023-02-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Viable Research Management_Site number 131, Phoenix, Arizona
  - Mayo Clinic - Scottsdale_Site number 150, Scottsdale, Arizona
  - University of California, SD_Site number 008, La Jolla, California
  - Pacific Arthrirtis Care Center_Site number 136, Los Angeles, California
  - University of California - Los Angeles_Site number 104, Los Angeles, California
  - Stanford University Medical Center_Site number 143, Palo Alto, California
  - University of Connecticut_Site number 147, Farmington, Connecticut
  - Yale University School of Medicine_Site number 140, New Haven, Connecticut
  - Georgetown University_Site number 035, Washington D.C., District of Columbia
  - St. Francis Medical_Site number 085, Clearwater, Florida
  - Omega Research Consultants_Site number 133, DeBary, Florida
  - Northwestern Medicine_Site number 124, Chicago, Illinois
  - DelRicht Research_Site number 159, New Orleans, Louisiana
  - Johns Hopkins University School of Medicine_Site number 134, Baltimore, Maryland
  - Massachusetts General Hospital_Site number 002, Boston, Massachusetts
  - Boston University_Site number 137, Boston, Massachusetts
  - University of Minnesota_Site number 051, Minneapolis, Minnesota
  - Mayo Clinic_Site number 146, Rochester, Minnesota
  - Hospital For Special Surgery_Site number 138, New York, New York
  - Columbia University Medical Center_Site number 086, New York, New York
  - Thomas Jefferson University Hospital_Site number 096, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center_Site number 149, Pittsburgh, Pennsylvania
  - Medical University of South Carolina_Site number 054, Charleston, South Carolina
  - Virginia Mason Medical Center_Site number 145, Seattle, Washington
  - Premier Clinical Research_Site number 130, Spokane, Washington
  - Froedtert Hospital and the Medical College of Wisconsin_Site number 012, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Derived] Chung L, Silver RM, Steen V, Furst DE, Castelino FV, Trojanowski M, Spiera R, Domsic R, Rodriguez-Pla A, Katsumoto TR, Goulaouic H, Wang H, Espinasse M, El-Chemaly S, Wang R. Belumosudil in diffuse cutaneous systemic sclerosis: a randomized, double-blind, open-label extension, placebo-controlled, phase 2 study. Rheumatology (Oxford). 2025 Jul 1;64(7):4299-4308. doi: 10.1093/rheumatology/keaf062. PMID 40088930

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 26 active sites in the United States. A total of 48 participants were screened from 26 June 2019 to 24 January 2022, of which 12 participants were screen failures. Screen failures were mainly due to not meeting eligibility criteria.
Pre-assignment Details: A total of 36 participants were enrolled and randomized into 3 groups in 1:1:1 ratio in double blind (DB) period of this study. The study was DB for first 28 weeks followed by an open-label extension (OLE) period of 24 weeks. After unblinding (i.e., in OLE), the participants who received belumosudil in DB period continued on same belumosudil dose whereas participants who received placebo were re-randomized in OLE period to one of the belumosudil doses (200 mg QD or 200 mg BID) in a 1:1 ratio.
Groups:
- Belumosudil QD/Belumosudil QD: Participants received belumosudil 200 milligrams (mg) tablet, once daily (QD) orally, for 28 weeks during the DB period. After completion of DB period, participants entered OLE period and continued to receive belumosudil 200 mg tablet QD orally for 24 weeks in OLE period (i.e., up to Week 52).
- Belumosudil BID/Belumosudil BID: Participants received belumosudil 200 mg tablet twice daily (BID) orally, for 28 weeks during the DB period. After completion of DB period, participants entered OLE period and continued to receive belumosudil 200 mg tablet BID orally for 24 weeks in OLE period (i.e., up to Week 52).
Period: DB Period (28 Weeks)
Arm/Group | Belumosudil QD/Belumosudil QD | Belumosudil BID/Belumosudil BID | DB Period: Placebo | OLE Period: Placebo/Belumosudil QD | OLE Period: Placebo/Belumosudil BID
Started | 12 | 12 | 12 | 0 | 0
Treated | 11 | 12 | 12 | 0 | 0
Completed | 10 | 10 | 11 | 0 | 0
Not Completed | 2 | 2 | 1 | 0 | 0
Not completed — Randomized not treated | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Period: OLE Period (24 Weeks)
Arm/Group | Belumosudil QD/Belumosudil QD | Belumosudil BID/Belumosudil BID | DB Period: Placebo | OLE Period: Placebo/Belumosudil QD | OLE Period: Placebo/Belumosudil BID
Started | 10 | 10 | 0 (Participants who completed DB period in this arm were re-randomized to 2 different arms Belumosudil (QD or BID) in OLE period.) | 5 (Participants who received placebo and completed DB period and were re-randomized to QD arm in the OLE period.) | 6 (Participants who received placebo and completed DB period and were re-randomized to BID arm in the OLE period.)
Completed | 10 | 7 | 0 | 5 | 6
Not Completed | 0 | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 0 | 0 | 0
Not completed — Other-unspecified | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on modified intent-to-treat (mITT) population which included all participants who received at least one dose of the study drug.
Groups:
- DB Period: Belumosudil QD: Participants received belumosudil 200 mg tablet, orally QD for 28 weeks during the DB period.
- DB Period: Belumosudil BID: Participants received belumosudil 200 mg tablet, orally BID for 28 weeks during the DB period.
- Total: Total of all reporting groups
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo | Total
Number analyzed (Participants) | 11 | 12 | 12 | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.7 (11.99) | 49.7 (15.80) | 46.3 (10.64) | 49.5 (12.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 10 | 26
  Male | 4 | 3 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 0 | 4
  White | 8 | 8 | 11 | 27
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1 | 2
Modified Rodnan Skin Score (mRSS) [Mean (Standard Deviation); unit: score on a scale] — Investigator assessed skin thickness by simple palpation on 17 different skin sites (e.g., face, hands, fingers; proximal area of arms, distal area of the arms, thorax, abdomen; proximal area of the legs, and distal area of the legs, feet). Each skin site was rated on 0 to 3 scale; where 0 = normal skin, 1 = mild, 2 = moderate, and 3 = severe thickness and unable to pinch. Individual skin site scores in 17 body areas were summed and defined as total mRSS which ranged from 0 (normal skin) to 51 (severe thickening), where higher score indicated more severity of skin thickening/worst outcome.
  score on a scale | 26.5 (6.47) | 25.2 (5.29) | 23.1 (4.85) | 24.9 (5.57)
Percent predicted forced vital capacity (FVC) [Mean (Standard Deviation); unit: percent predicted FVC] — FVC was the total amount of air exhaled from the lungs during the lung function test measured by spirometer which assessed the change in lung function related to the disease status of an underlying interstitial lung disease.
  percent predicted FVC | 98.6 (15.91) | 84.0 (15.90) | 86.2 (17.75) | 89.3 (17.32)
Physician Global Assessment of Participant's Overall Health Using Visual Analogue Scale (VAS) Score [Mean (Standard Deviation); unit: score on a scale] — The Physician Global Assessment (reported by the physician) quantified the participant's overall health during the last week based on VAS which ranged from 0 (extremely poor) to 100 (excellent). Higher score indicated better outcome.
  score on a scale | 43.1 (17.89) | 58.2 (12.59) | 43.0 (18.06) | 48.2 (17.43)
Patient Global Assessment of Participant's Overall Health Using VAS Score [Mean (Standard Deviation); unit: score on a scale] — The Patient Global Assessment (reported by participant) quantified the participant's overall health during the last week based on a VAS which ranged from 0 (extremely poor) to 100 (excellent). Higher score indicated better outcome.
  score on a scale | 56.5 (22.47) | 58.6 (16.92) | 59.6 (16.72) | 58.3 (18.26)
Scleroderma Health Assessment Questionnaire-Disability Index (SHAQ-DI) Total Score [Mean (Standard Deviation); unit: score on a scale] — SHAQ-DI included general HAD-DI assessment and 6 scleroderma-specific VAS items. HAD-DI included 8 domains addressing scleroderma related manifestations that contribute to disability. For each question, level of difficulty was scored from 0 to 3, where 0=no difficulty, 1=some difficulty, 2=much difficulty, 3=unable to do. Some domains in SHAQ are VAS that were measured first and then changed to 0-3 scale. SHAQ-DI total score=sum of domain scores divided by number of domains answered, ranged 0 (no difficulty) to 3 (maximum difficulty), where higher score=greater disability/worse functionality.
  score on a scale | 1.489 (0.719) | 1.396 (0.626) | 1.302 (0.712) | 1.393 (0.670)

OUTCOME MEASURES:

1. Primary Outcome: DB Period: Number of Participants With Combined Response Index in Diffuse Cutaneous Systemic Sclerosis (CRISS) Score Greater Than or Equal to (>=) 60 Percent (%) at Week 24
Description: CRISS components included the following domains: mRSS, FVC percent predicted, physician global assessment, patient global assessment, and SHAQ-DI. An algorithm determines the predicted probability of improvement from Baseline by incorporating change from baseline in the mRSS, FVC percent predicted, physician and patient global assessments, and SHAQ-DI. The outcome is a continuous variable between 0.0 and 1.0 (0 to 100%). Higher score indicated greater probability of improvement. CRISS score >= 60% was considered the minimally important difference. Participants were not considered improved and assigned a probability of improving equal to 0.0 if they developed new onset of renal crisis, new onset or worsening of lung fibrosis, new onset of pulmonary arterial hypertension, or new onset of left ventricular failure during the trial. Last observation carried forward (LOCF) method was used to handle missing data.
Time Frame: Week 24
Population: Analysis was performed on mITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 11 | 12 | 12
Participants | 6 | 3 | 7
Statistical Analysis 1: Comparison: DB Period: Belumosudil QD vs DB Period: Placebo; Belumosudil 200 mg QD versus Placebo; Test type: Superiority — The LOCF imputation was followed by logistic regression analysis. Comparison analysis between belumosudil dose regimen and placebo was performed using a logistic regression analysis with treatment in the model; p = 0.9472, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 1.06, 95% CI 2-sided [0.19 to 5.82]
Statistical Analysis 2: Comparison: DB Period: Belumosudil BID vs DB Period: Placebo; Belumosudil 200 mg BID versus Placebo; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.3078, Regression, Logistic — Threshold for significance at 0.05 level; Odds Ratio (OR) = 0.39, 95% CI 2-sided [0.07 to 2.35]

2. Secondary Outcome: DB Period: Combined Response Index in Diffuse Cutaneous Systemic Sclerosis Score at Week 24
Description: CRISS components included the following domains: mRSS, FVC percent predicted, physician global assessment, patient global assessment, and SHAQ-DI. An algorithm determines the predicted probability of improvement from Baseline by incorporating change from baseline in the mRSS, FVC percent predicted, physician and patient global assessments, and SHAQ-DI. The outcome is a continuous variable between 0.0 and 1.0 (0 to 100%). A higher score indicated greater probability of improvement. Participants were not considered improved and assigned a probability of improving equal to 0.0 if they developed new onset of renal crisis, new onset or worsening of lung fibrosis, new onset of pulmonary arterial hypertension, new onset of left ventricular failure during the trial. Least squares (LS) mean and 95% confidence interval (CI) were obtained by mixed-effect model for repeated measures (MMRM).
Time Frame: Week 24
Population: Analysis was performed on mITT population. LOCF method was used to handle missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 11 | 12 | 12
score on a scale | 14.30 [9.47 to 19.12] | 10.16 [5.41 to 14.91] | 14.34 [10.04 to 18.64]
Statistical Analysis 1: Comparison: DB Period: Belumosudil QD vs DB Period: Placebo; Belumosudil 200 mg QD versus Placebo; Test type: Superiority — MMRM analysis used rank-transformed data, with CRISS score as a dependent variable and treatment, visit, and visit x treatment interaction as fixed effects. Visit was a repeated factor, and analyses were done through week 24; p = 0.9889, MMRM — Threshold for significance at 0.05 level; Least square mean difference = -0.04, 95% CI 2-sided [-6.51 to 6.42]
Statistical Analysis 2: Comparison: DB Period: Belumosudil BID vs DB Period: Placebo; Belumosudil 200 mg BID versus Placebo; Test type: Superiority — MMRM analysis using rank-transformed data, with CRISS score as a dependent variable and treatment, visit, and visit x treatment interaction as fixed effects. Visit was a repeated factor, and analyses were done through week 24; p = 0.1916, MMRM — Threshold for significance at 0.05 level; Least square mean difference = -4.18, 95% CI 2-sided [-10.59 to 2.23]

3. Secondary Outcome: OLE Period: Combined Response Index in Diffuse Cutaneous Systemic Sclerosis Score at Week 52
Description: CRISS components included following domains: mRSS, percent predicted FVC, physician global assessment, patient global assessment, and SHAQ-DI. An algorithm determines the predicted probability of improvement from Baseline by incorporating change from baseline in the mRSS, FVC percent predicted, physician and patient global assessments, and SHAQ-DI. The outcome was a continuous variable between 0.0 and 1.0 (0 to 100%). Higher score indicated greater probability of improvement. Participants were not considered improved and assigned a probability of improving equal to 0.0 if they developed new onset of renal crisis, new onset or worsening of lung fibrosis, new onset of pulmonary arterial hypertension, new onset of left ventricular failure during the trial. LOCF method was used to handle missing data.
Time Frame: Week 52
Population: Analysis was performed on mITT population.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- OLE Period: Belumosudil QD: Participants who had received belumosudil QD in the DB period continued to receive belumosudil 200 mg tablet QD orally for 24 weeks in OLE period (i.e., up to Week 52).
- OLE Period: Belumosudil BID: Participants who had received belumosudil BID in the DB period continued to receive belumosudil 200 mg tablet BID orally for 24 weeks in OLE period (i.e., up to Week 52).
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 10 | 5 | 10 | 6
score on a scale | 87.46 (27.376) | 7.16 (8.749) | 64.37 (41.950) | 11.62 (19.282)

4. Secondary Outcome: DB Period: Change From Baseline in Modified Rodnan Skin Score (mRSS) at Week 24
Description: mRSS is an accepted clinical measure of skin thickness. The investigator assessed the skin thickness using the mRSS through simple palpation on 17 different skin sites (e.g., face, hands, fingers; proximal area of the arms, distal area of the arms, thorax, abdomen; proximal area of the legs, and distal area of the legs, feet). Each skin site was rated on a 0 to 3 scale; where 0 = normal skin, 1 = mild thickness, 2 = moderate thickness, and 3 = severe thickness and unable to pinch. Individual site skin scores in the 17 body areas were summed and defined as the total mRSS which ranged from 0 (normal skin) to 51 (severe thickening), where higher score indicated more severity of skin thickening/worst outcome. LS mean and 95% CI were calculated using MMRM model.
Time Frame: Baseline, Week 24
Population: Analysis was performed on mITT population. For participants who received placebo/belumosudil in the DB period, the Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in the DB period.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 11 | 12 | 12
score on a scale | -9.2 [-12.2 to -6.2] | -4.0 [-7.0 to -1.0] | -8.6 [-11.4 to -5.8]
Statistical Analysis 1: Comparison: DB Period: Belumosudil QD vs DB Period: Placebo; Belumosudil 200 mg QD versus Placebo; Test type: Superiority; p = 0.7710, MMRM — Threshold for significance at 0.05 level; Least square mean difference = -0.6, 95% CI 2-sided [-4.7 to 3.6]
Statistical Analysis 2: Comparison: DB Period: Belumosudil BID vs DB Period: Placebo; Belumosudil 200 mg BID versus Placebo; Test type: Superiority; p = 0.0308, MMRM — Threshold for significance at 0.05 level; Least square mean difference = 4.6, 95% CI 2-sided [0.5 to 8.8]

5. Secondary Outcome: DB Period: Change From Baseline in Percent Predicted Forced Vital Capacity (FVC) at Week 24
Description: FVC was the total amount of air exhaled from the lungs during the lung function test measured by spirometer which assessed the change in lung function related to the disease status of an underlying interstitial lung disease (ILD). LS mean and 95% CI were obtained from MMRM model.
Time Frame: Baseline, Week 24
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percent predicted FVC
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 11 | 12 | 12
percent predicted FVC | 0.6 [-4.0 to 5.2] | -2.3 [-7.2 to 2.5] | -0.8 [-5.2 to 3.6]
Statistical Analysis 1: Comparison: DB Period: Belumosudil QD vs DB Period: Placebo; Belumosudil 200 mg QD versus Placebo; Test type: Superiority; p = 0.6533, MMRM — Threshold for significance at 0.05 level; Least square mean difference = 1.4, 95% CI 2-sided [-4.9 to 7.7]
Statistical Analysis 2: Comparison: DB Period: Belumosudil BID vs DB Period: Placebo; Belumosudil 200 mg BID versus Placebo; Test type: Superiority; p = 0.6338, MMRM — Threshold for significance at 0.05 level; Least square mean difference = -1.5, 95% CI 2-sided [-8.1 to 5.0]

6. Secondary Outcome: DB Period: Change From Baseline in Physician Global Assessment of Participant's Overall Health Using Visual Analogue Scale Score at Week 24
Description: The Physician Global Assessment (reported by the physician) quantified the participant's overall health during the last week based on VAS which ranged from 0 (extremely poor) to 100 (excellent). Higher score indicated better outcome. LS mean and 95% CI were obtained from MMRM model.
Time Frame: Baseline, Week 24
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 11 | 12 | 12
score on a scale | 22.4 [10.0 to 34.8] | -0.8 [-13.2 to 11.6] | 7.8 [-4.1 to 19.6]
Statistical Analysis 1: Comparison: DB Period: Belumosudil QD vs DB Period: Placebo; Belumosudil 200 mg QD versus Placebo; Test type: Superiority; p = 0.0916, MMRM — Threshold for significance at 0.05 level; Least square mean difference = 14.6, 95% CI 2-sided [-2.5 to 31.8]
Statistical Analysis 2: Comparison: DB Period: Belumosudil BID vs DB Period: Placebo; Belumosudil 200 mg BID versus Placebo; Test type: Superiority; p = 0.3146, MMRM; Least square mean difference = -8.6, 95% CI 2-sided [-25.7 to 8.6]

7. Secondary Outcome: DB Period: Change From Baseline in Patient Global Assessment of Participant's Overall Health Using Visual Analogue Scale Score at Week 24
Description: The Patient Global Assessment (reported by participant) quantified the participant's overall health during the last week based on a VAS which ranged from 0 (extremely poor) to 100 (excellent). Higher score indicated better outcome. LS mean and 95% CI were obtained from MMRM model.
Time Frame: Baseline, Week 24
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 11 | 12 | 12
score on a scale | -5.8 [-22.4 to 10.8] | 3.5 [-13.1 to 20.1] | 4.2 [-11.4 to 19.8]
Statistical Analysis 1: Comparison: DB Period: Belumosudil QD vs DB Period: Placebo; Belumosudil 200 mg QD versus Placebo; Test type: Superiority; p = 0.3753, MMRM — Threshold for significance at 0.05 level; Least square mean difference = -10.0, 95% CI 2-sided [-32.8 to 12.8]
Statistical Analysis 2: Comparison: DB Period: Belumosudil BID vs DB Period: Placebo; Belumosudil 200 mg BID versus Placebo; Test type: Superiority; p = 0.9481, MMRM — Threshold for significance at 0.05 level; Least square mean difference = -0.7, 95% CI 2-sided [-23.5 to 22.1]

8. Secondary Outcome: DB Period: Change From Baseline in Scleroderma Health Assessment Questionnaire-Disability Index (SHAQ-DI) Total Score at Week 24
Description: SHAQ-DI included the general health assessment questionnaire-disability index (HAD-DI) assessment and 6 scleroderma-specific VAS items to explore impact of participant's disease. General HAD-DI assessment included 8 domains: dressing, arising, eating, walking, hygiene, reach, grip, and activities addressing scleroderma related manifestations that contribute to disability. It is a quality of life measure. For each question, level of difficulty was scored from 0 to 3, where 0=no difficulty, 1=some difficulty, 2=much difficulty, 3=unable to do. Some domains in the SHAQ are visual analog scales that are measured first and then changed to a 0-3 scale. SHAQ-DI total score was computed as the sum of domain scores divided by the number of domains answered and it ranged from 0 (no difficulty) to 3 (maximum difficulty), where higher score indicated greater disability/worse functionality. LS mean and 95% CI were obtained from MMRM model.
Time Frame: Baseline, Week 24
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 11 | 12 | 12
score on a scale | -0.187 [-0.449 to 0.074] | -0.112 [-0.374 to 0.149] | -0.152 [-0.393 to 0.090]
Statistical Analysis 1: Comparison: DB Period: Belumosudil QD vs DB Period: Placebo; Belumosudil 200 mg QD versus Placebo; Test type: Superiority; p = 0.8387, MMRM — Threshold for significance at 0.05 level; Least square mean difference = -0.036, 95% CI 2-sided [-0.392 to 0.320]
Statistical Analysis 2: Comparison: DB Period: Belumosudil BID vs DB Period: Placebo; Belumosudil 200 mg BID versus Placebo; Test type: Superiority; p = 0.8234, MMRM — Threshold for significance at 0.05 level; Least square mean difference = 0.039, 95% CI 2-sided [-0.317 to 0.395]

9. Secondary Outcome: DB Period: Percentage Improvement in Modified Rodnan Skin Score at Week 24
Description: The mRSS is an accepted clinical measure of skin thickness. The investigator assessed the skin thickness using the mRSS through simple palpation on 17 different skin sites (e.g., face, hands, fingers; proximal area of the arms, distal area of the arms, thorax, abdomen; proximal area of the legs, and distal area of the legs, feet). Each skin site was rated on 0 to 3 scale; where 0 = normal skin, 1 = mild thickness, 2 = moderate thickness, and 3 = severe thickness and unable to pinch. Individual site skin scores in the 17 body areas were summed and defined as the total mRSS which ranged from 0 (normal skin) to 51 (severe thickening), where higher score indicated more severity of skin thickening/worst outcome. Percentage improvement = change from Baseline value divided by Baseline value*100. LS mean and 95% CI were obtained from MMRM model.
Time Frame: Baseline, Week 24
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage improvement
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 11 | 12 | 12
percentage improvement | 37.268 [23.074 to 51.462] | 19.262 [5.068 to 33.457] | 40.277 [27.047 to 53.507]
Statistical Analysis 1: Comparison: DB Period: Belumosudil QD vs DB Period: Placebo; Belumosudil 200 mg QD versus Placebo; Test type: Superiority; p = 0.7535, MMRM — Threshold for significance at 0.05 level; Least square mean difference = -3.009, 95% CI 2-sided [-22.413 to 16.395]
Statistical Analysis 2: Comparison: DB Period: Belumosudil BID vs DB Period: Placebo; Belumosudil 200 mg BID versus Placebo; Test type: Superiority; p = 0.0348, MMRM — Threshold for significance at 0.05 level; Least square mean difference = -21.015, 95% CI 2-sided [-40.419 to -1.611]

10. Secondary Outcome: DB Period: Percentage Improvement in Physician Global Assessment of Participant's Overall Health Using Visual Analogue Scale (VAS) Score at Week 24
Description: The Physician Global Assessment (reported by the physician) quantified the participant's overall health during the last week based on VAS which ranged from 0 (extremely poor) to 100 (excellent). Higher score indicated better outcome. Percentage improvement = change from Baseline value divided by Baseline value*100. LS mean and 95% CI were obtained from MMRM model.
Time Frame: Baseline, Week 24
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage improvement
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 11 | 12 | 12
percentage improvement | 68.790 [38.465 to 99.115] | 1.240 [-29.085 to 31.564] | 23.224 [-5.757 to 52.204]
Statistical Analysis 1: Comparison: DB Period: Belumosudil QD vs DB Period: Placebo; Belumosudil 200 mg QD versus Placebo; Test type: Superiority; p = 0.0343, MMRM — Threshold for significance at 0.05 level; Least square mean difference = 45.566, 95% CI 2-sided [3.621 to 87.512]
Statistical Analysis 2: Comparison: DB Period: Belumosudil BID vs DB Period: Placebo; Belumosudil 200 mg BID versus Placebo; Test type: Superiority; p = 0.2922, MMRM — Threshold for significance at 0.05 level; Least square mean difference = -21.984, 95% CI 2-sided [-63.930 to 19.962]

11. Secondary Outcome: DB Period: Percentage Improvement in Patient Global Assessment of Participant's Overall Health Using Visual Analogue Scale Score at Week 24
Description: The Patient Global Assessment (reported by participant) quantified the participant's overall health during the last week based on a VAS which ranged from 0 (extremely poor) to 100 (excellent). Higher score indicated better outcome. Percentage improvement = change from Baseline value divided by Baseline value*100. LS mean and 95% CI were obtained from MMRM model.
Time Frame: Baseline, Week 24
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage improvement
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 11 | 12 | 12
percentage improvement | -2.583 [-42.146 to 36.981] | 18.194 [-21.369 to 57.758] | 14.174 [-22.838 to 51.186]
Statistical Analysis 1: Comparison: DB Period: Belumosudil QD vs DB Period: Placebo; Belumosudil 200 mg QD versus Placebo; Test type: Superiority; p = 0.5320, MMRM — Threshold for significance at 0.05 level; Least square mean difference = -16.757, 95% CI 2-sided [-70.933 to 37.419]
Statistical Analysis 2: Comparison: DB Period: Belumosudil BID vs DB Period: Placebo; Belumosudil 200 mg BID versus Placebo; Test type: Superiority; p = 0.8804, MMRM — Threshold for significance at 0.05 level; Least square mean difference = 4.020, 95% CI 2-sided [-50.156 to 58.196]

12. Secondary Outcome: DB Period: Percentage Improvement in Scleroderma Health Assessment Questionnaire-Disability Index (SHAQ-DI) Total Score at Week 24
Description: SHAQ-DI included general HAD-DI assessment and 6 scleroderma-specific VAS items to explore impact of participant's disease. General HAD-DI assessment included 8 domains: dressing, arising, eating, walking, hygiene, reach, grip, and activities addressing scleroderma related manifestations that contribute to disability. For each question, level of difficulty was scored from 0 to 3, where 0=no difficulty, 1=some difficulty, 2=much difficulty, 3=unable to do. Some domains in SHAQ are visual analog scales that are measured first and then changed to 0-3 scale. SHAQ-DI total score was computed as sum of domain scores divided by number of domains answered and it ranged from 0 (no difficulty) to 3 (maximum difficulty), where higher score indicated greater disability/worse functionality. Percentage improvement = change from Baseline value divided by Baseline value*100. LS mean and 95% CI were obtained from MMRM model.
Time Frame: Baseline, Week 24
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage improvement
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 11 | 12 | 12
percentage improvement | 12.065 [-54.683 to 78.813] | -37.898 [-101.221 to 25.424] | 4.544 [-53.353 to 62.440]
Statistical Analysis 1: Comparison: DB Period: Belumosudil QD vs DB Period: Placebo; Belumosudil 200 mg QD versus Placebo; Test type: Superiority; p = 0.8628, MMRM — Threshold for significance at 0.05 level; Least square mean difference = 7.522, 95% CI 2-sided [-80.837 to 95.880]
Statistical Analysis 2: Comparison: DB Period: Belumosudil BID vs DB Period: Placebo; Belumosudil 200 mg BID versus Placebo; Test type: Superiority; p = 0.3196, MMRM; Least square mean difference = -42.442, 95% CI 2-sided [-128.242 to 43.359]

13. Secondary Outcome: OLE Period: Change From Baseline in Modified Rodnan Skin Score at Week 52
Description: The mRSS is an accepted clinical measure of skin thickness. The investigator assessed the skin thickness using the mRSS through simple palpation on 17 different skin sites (e.g., face, hands, fingers; proximal area of the arms, distal area of the arms, thorax, abdomen; proximal area of the legs, and distal area of the legs, feet). Each skin site was rated on a 0 to 3 scale; where 0 = normal skin, 1 = mild thickness, 2 = moderate thickness, and 3 = severe thickness and unable to pinch. Individual site skin scores in the 17 body areas were summed and defined as the total mRSS which ranged from 0 (normal skin) to 51 (severe thickening), where higher score indicated more severity of skin thickening/worst outcome. In the below data table, 'number analyzed' = participants with available data for each specified category.
Time Frame: Baseline, Week 52
Population: Analyzed on mITT. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 10 | 5 | 10 | 6
score on a scale
  Baseline | 25.7 (6.15) | 12.8 (9.91) | 24.0 (4.81) | 14.7 (5.75)
  Change at Week 52: number analyzed (Participants) | 10 | 5 | 7 | 6
  Change at Week 52 | -14.4 (4.09) | -2.0 (5.10) | -9.4 (3.51) | -2.5 (1.64)

14. Secondary Outcome: OLE Period: Change From Baseline in Percent Predicted Forced Vital Capacity at Week 52
Description: FVC was the total amount of air exhaled from the lungs during the lung function test measured by spirometer which assessed the change in lung function related to the disease status of an underlying ILD. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period.
Time Frame: Baseline, Week 52
Population: Analysis was performed on mITT population. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: percent predicted FVC
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 10 | 5 | 10 | 6
percent predicted FVC
  Baseline | 98.5 (16.77) | 95.8 (11.26) | 83.3 (17.47) | 76.7 (18.42)
  Change at Week 52: number analyzed (Participants) | 10 | 5 | 6 | 6
  Change at Week 52 | -4.1 (5.36) | 1.0 (6.71) | -0.7 (13.69) | 2.7 (4.18)

15. Secondary Outcome: OLE Period: Change From Baseline in Physician Global Assessment of Participant's Overall Health Using Visual Analogue Scale (VAS) Score at Week 52
Description: The Physician Global Assessment (reported by the physician) quantified the participant's overall health during the last week based on VAS which ranged from 0 (extremely poor) to 100 (excellent). Higher score indicated better outcome. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period.
Time Frame: Baseline, Week 52
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 10 | 5 | 10 | 6
score on a scale
  Baseline | 41.5 (18.02) | 60.6 (20.66) | 59.7 (12.87) | 43.3 (25.07)
  Change at Week 52: number analyzed (Participants) | 10 | 5 | 7 | 6
  Change at Week 52 | 22.2 (27.80) | -6.2 (18.51) | 7.0 (29.58) | 3.3 (17.45)

16. Secondary Outcome: OLE Period: Change From Baseline in Patient Global Assessment of Participant's Overall Health Using Visual Analogue Scale Score at Week 52
Description: The Patient Global Assessment (reported by participant) quantified the participant's overall health during the last week based on a VAS which ranged from 0 (extremely poor) to 100 (excellent). Higher score indicated better outcome. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period.
Time Frame: Baseline, Week 52
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 10 | 5 | 10 | 6
score on a scale
  Baseline | 61.1 (17.24) | 51.8 (26.85) | 57.6 (18.50) | 43.7 (20.72)
  Change at Week 52: number analyzed (Participants) | 10 | 5 | 7 | 6
  Change at Week 52 | -12.1 (30.58) | 15.0 (29.91) | -2.4 (13.82) | 16.2 (33.91)

17. Secondary Outcome: OLE Period: Change From Baseline in Scleroderma Health Assessment Questionnaire-Disability Index Total Score at Week 52
Description: SHAQ-DI included general HAD-DI assessment and 6 scleroderma-specific VAS items to explore the impact of participant's disease. General HAD-DI assessment included 8 domains: dressing, arising, eating, walking, hygiene, reach, grip, and activities addressing scleroderma related manifestations that contribute to disability. For each question, level of difficulty was scored from 0 to 3, where 0=no difficulty, 1=some difficulty, 2=much difficulty, 3=unable to do. Some domains in SHAQ are visual analog scales that are measured first and then changed to a 0-3 scale. SHAQ-DI total score was computed as sum of domain scores divided by the number of domains answered and it ranged from 0 (no difficulty) to 3 (maximum difficulty), where higher score indicated greater disability/worse functionality. In the data table below, 'number analyzed' = participants with available data for each specified category.
Time Frame: Baseline, Week 52
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 10 | 5 | 10 | 6
score on a scale
  Baseline | 1.513 (0.753) | 1.275 (0.582) | 1.388 (0.686) | 1.042 (0.727)
  Change at Week 52: number analyzed (Participants) | 10 | 5 | 7 | 6
  Change at Week 52 | -0.200 (0.422) | -0.050 (0.068) | -0.089 (0.312) | 0.063 (0.172)

18. Secondary Outcome: OLE Period: Percentage Improvement in Modified Rodnan Skin Score at Week 52
Description: The mRSS is an accepted clinical measure of skin thickness. The investigator assessed the skin thickness using the mRSS through simple palpation on 17 different skin sites in (e.g., face, hands, fingers; proximal area of the arms, distal area of the arms, thorax, abdomen; proximal area of the legs, and distal area of the legs, feet). Each skin site was rated on a 0 to 3 scale; where 0 = normal skin, 1 = mild thickness, 2 = moderate thickness, and 3 = severe thickness and unable to pinch. Individual site skin scores in the 17 body areas were summed and defined as the total mRSS which ranged from 0 (normal skin) to 51 (severe thickening), where higher score indicated more severity of skin thickening/worst outcome. Percentage improvement = change from Baseline value divided by Baseline value*100. In the data table below, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Time Frame: Baseline, Week 52
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percentage improvement
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 10 | 5 | 7 | 6
percentage improvement | 57.119 (13.719) | -13.687 (76.463) | 41.123 (16.813) | 20.959 (14.344)

19. Secondary Outcome: OLE Period: Percentage Improvement Physician Global Assessment of Participant's Overall Health Using Visual Analogue Scale (VAS) Score at Week 52
Description: The Physician Global Assessment (reported by the physician) quantified the participant's overall health during the last week based on VAS which ranged from 0 (extremely poor) to 100 (excellent). Higher score indicated better outcome. Percentage improvement = change from Baseline value divided by Baseline value*100. In the data below, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Time Frame: Baseline, Week 52
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percentage improvement
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 10 | 5 | 7 | 6
percentage improvement | 76.075 (73.169) | -8.138 (29.916) | 22.014 (56.885) | 24.287 (71.494)

20. Secondary Outcome: OLE Period: Percentage Improvement in Patient Global Assessment of Participant's Overall Health Using Visual Analogue Scale Score at Week 52
Description: The Patient Global Assessment (reported by participant) quantified the participant's overall health during the last week based on a VAS which ranged from 0 (extremely poor) to 100 (excellent). Higher score indicated better outcome. Percentage improvement = change from Baseline value divided by Baseline value*100. In the data table below, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Time Frame: Baseline, Week 52
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percentage improvement
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 10 | 5 | 7 | 6
percentage improvement | -7.833 (57.154) | 40.966 (82.168) | -3.797 (26.577) | 79.771 (122.523)

21. Secondary Outcome: OLE Period: Percentage Improvement in Scleroderma Health Assessment Questionnaire-Disability Index Score at Week 52
Description: SHAQ-DI: general health assessment questionnaire-disability index (HAD-DI) assessment and 6 scleroderma-specific VAS items to explore impact of participant's disease. General HAD-DI assessment included 8 domains: dressing, arising, eating, walking, hygiene, reach, grip, and activities addressing scleroderma related manifestations that contribute to disability. For each question, level of difficulty was scored from 0 to 3; 0=no difficulty, 1=some difficulty, 2=much difficulty, 3=unable to do. Some domains in SHAQ are visual analog scales that are measured first and then changed to 0-3 scale. SHAQ-DI total score computed as sum of domain scores divided by number of domains answered ranging 0 (no difficulty) to 3 (maximum difficulty), where higher score indicated greater disability/worse functionality. Percentage improvement = change from Baseline value divided by Baseline value*100. 'overall number of participants analyzed' = participants with available data for this outcome measure.
Time Frame: Baseline, Week 52
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: percentage improvement
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 9 | 5 | 7 | 6
percentage improvement | 15.496 (33.762) | 5.667 (8.788) | -33.254 (118.780) | -15.347 (35.326)

22. Secondary Outcome: DB Period: Change From Baseline in Percent Predicted Forced Vital Capacity Level at Week 24-ILD Participants
Description: FVC was the total amount of air exhaled from the lungs during the lung function test measured by spirometer which assessed the change in lung function related to the disease status of an underlying ILD. For participants who received placebo/belumosudil in the DB period, the Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in the DB period. Change from Baseline in percent predicted FVC level at Week 24 in participants with ILD is reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: Analysis was performed on participants with ILD. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: percent predicted FVC
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 4 | 7 | 6
percent predicted FVC
  Baseline | 93.3 (13.15) | 81.3 (15.77) | 80.2 (19.79)
  Change at Week 24: number analyzed (Participants) | 4 | 5 | 5
  Change at Week 24 | -2.3 (15.73) | -2.2 (5.45) | 0.4 (2.79)

23. Secondary Outcome: DB Period: Change From Baseline in Percent Predicted Diffusing Capacity of the Lungs for Carbon Monoxide (DLco) at Week 24-ILD Participants
Description: DLco is a measurement of the ability of the lungs to transfer gases from the air to the blood. Participants breathe in (inhale) air containing a very small, harmless amount of a tracer gas, such as carbon monoxide. Participants hold their breath for 10 seconds, then rapidly blow it out (exhale). The exhaled gas was tested to determine amount of the tracer gas absorbed during the breath. For participants who received placebo/belumosudil in the DB period, the Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in the DB period. Change from Baseline in percent predicted DLco at Week 24 in participants with ILD is reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: percent predicted DLco
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 4 | 6 | 4
percent predicted DLco
  Baseline | 76.3 (20.45) | 60.3 (15.98) | 60.5 (10.21)
  Change at Week 24: number analyzed (Participants) | 3 | 5 | 3
  Change at Week 24 | -6.3 (10.21) | 4.4 (7.47) | 1.3 (4.16)

24. Secondary Outcome: DB Period: Change From Baseline in Percent Predicted Forced Expiratory Volume (FEV1) at Week 24-ILD Participants
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by a spirometer. For participants who received placebo/belumosudil in the DB period, the Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in the DB period. Change from Baseline in percent predicted FEV1 at Week 24 in participants with ILD is reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: percent predicted FEV1
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 4 | 7 | 5
percent predicted FEV1
  Baseline | 95.3 (7.37) | 83.1 (14.88) | 86.4 (17.29)
  Change at Week 24: number analyzed (Participants) | 3 | 5 | 4
  Change at Week 24 | -8.7 (12.22) | -2.2 (6.02) | 0.8 (2.75)

25. Secondary Outcome: DB Period: Change From Baseline in Percent Predicted Residual Volume (RV) at Week 24-ILD Participants
Description: RV is the volume of air remaining in the lungs after maximum forceful expiration. For participants who received placebo/belumosudil in the DB period, the Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in the DB period. Change from Baseline in percent predicted RV at Week 24 in participants with ILD is reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: percent predicted RV
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 3 | 7 | 5
percent predicted RV
  Baseline | 80.7 (26.58) | 73.7 (24.37) | 69.8 (27.97)
  Change at Week 24: number analyzed (Participants) | 3 | 5 | 4
  Change at Week 24 | -17.7 (8.96) | 0.2 (16.60) | 29.5 (18.08)

26. Secondary Outcome: DB Period: Change From Baseline in Percent Predicted Total Lung Capacity (TLC) at Week 24-ILD Participants
Description: TLC is the volume of air in the lungs upon the maximum effort of inspiration. For participants who received placebo/belumosudil in the DB period, the Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in the DB period. Change from Baseline in percent predicted TLC at Week 24 in participants with ILD is reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: percent predicted TLC
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 3 | 7 | 5
percent predicted TLC
  Baseline | 89.0 (18.03) | 79.0 (15.83) | 80.6 (19.71)
  Change at Week 24: number analyzed (Participants) | 3 | 5 | 4
  Change at Week 24 | -11.3 (4.62) | -2.2 (4.02) | 10.5 (7.05)

27. Secondary Outcome: OLE Period: Change From Baseline in Percent Predicted Forced Vital Capacity at Week 52-ILD Participants
Description: FVC was the total amount of air exhaled from the lungs during the lung function test measured by spirometer which assessed the change in lung function related to the disease status of an underlying ILD. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period. Change from Baseline in percent predicted FVC at Week 52 in participants with ILD is reported in this outcome measure.
Time Frame: Baseline, Week 52
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: percent predicted FVC
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 4 | 2 | 6 | 3
percent predicted FVC
  Baseline | 93.3 (13.15) | 97.5 (16.26) | 80.5 (17.12) | 68.0 (20.66)
  Change at Week 52: number analyzed (Participants) | 4 | 2 | 3 | 3
  Change at Week 52 | -7.3 (3.59) | -4.0 (2.83) | 3.7 (12.50) | 4.0 (5.29)

28. Secondary Outcome: OLE Period: Change From Baseline in Percent Predicted Diffusing Capacity of the Lungs for Carbon Monoxide at Week 52-ILD Participants
Description: DLco is a measurement of the ability of the lungs to transfer gases from the air to the blood. Participants breathe in (inhale) air containing a very small, harmless amount of a tracer gas, such as carbon monoxide. Participants hold their breath for 10 seconds, then rapidly blow it out (exhale). The exhaled gas was tested to determine amount of the tracer gas absorbed during the breath. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period. Change from Baseline in percent predicted DLco at Week 52 in participants with ILD is reported in this outcome measure.
Time Frame: Baseline, Week 52
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: percent predicted DLco
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 4 | 2 | 6 | 3
percent predicted DLco
  Baseline | 76.3 (20.45) | 78.0 (7.07) | 60.3 (15.98) | 56.3 (2.08)
  Change at Week 52: number analyzed (Participants) | 4 | 2 | 3 | 3
  Change at Week 52 | -9.0 (9.27) | 2.0 (7.07) | 6.0 (7.21) | 1.7 (11.72)

29. Secondary Outcome: OLE Period: Change From Baseline in Percent Predicted Forced Expiratory Volume at Week 52-ILD Participants
Description: FEV1 was the volume of air exhaled in the first second of a forced expiration as measured by a spirometer. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period. Change from Baseline in percent predicted FEV1 at Week 52 in participants with ILD is reported in this outcome measure.
Time Frame: Baseline, Week 52
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: percent predicted FEV1
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 4 | 2 | 6 | 3
percent predicted FEV1
  Baseline | 95.3 (7.37) | 101.5 (13.44) | 81.0 (15.07) | 70.0 (19.00)
  Change at Week 52: number analyzed (Participants) | 4 | 2 | 3 | 3
  Change at Week 52 | -6.8 (2.06) | -2.0 (4.24) | 4.0 (14.18) | -0.7 (7.09)

30. Secondary Outcome: OLE Period: Change From Baseline in Percent Predicted Residual Volume at Week 52-ILD Participants
Description: RV is the volume of air remaining in the lungs after maximum forceful expiration. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period. Change from Baseline in percent predicted RV at Week 52 in participants with ILD is reported in this outcome measure.
Time Frame: Baseline, Week 52
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: percent predicted RV
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 3 | 2 | 6 | 3
percent predicted RV
  Baseline | 80.7 (26.58) | 113.0 (36.77) | 76.2 (25.73) | 81.7 (31.66)
  Change at Week 52: number analyzed (Participants) | 3 | 2 | 3 | 2
  Change at Week 52 | -21.3 (22.50) | -28.0 (35.36) | 3.7 (11.93) | -22.5 (7.78)

31. Secondary Outcome: OLE Period: Change From Baseline in Percent Predicted Total Lung Capacity at Week 52-ILD Participants
Description: TLC is the volume of air in the lungs upon the maximum effort of inspiration. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period. Change from Baseline in percent predicted TLC at Week 52 in participants with ILD is reported in this outcome measure.
Time Frame: Baseline, Week 52
Population: as for outcome 22
Measure: Mean (Standard Deviation); unit: percent predicted TLC
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 3 | 2 | 6 | 3
percent predicted TLC
  Baseline | 89.0 (18.03) | 104.0 (14.14) | 79.7 (17.24) | 80.7 (19.14)
  Change at Week 52: number analyzed (Participants) | 3 | 2 | 3 | 2
  Change at Week 52 | -13.0 (11.14) | -10.0 (8.49) | 3.3 (3.06) | -11.0 (4.24)

32. Secondary Outcome: DB Period: Number of Participants With Lung Fibrosis at Baseline and Week 24-ILD Participants
Description: Lung fibrosis is a lung disease in which lung tissue becomes damaged and scared. Lung fibrosis was assessed using high-resolution computerized tomography (HRCT). HRCT is a type of computed tomography used to diagnose and stage the severity. Pure ground-class opacity, pulmonary fibrosis and honeycombing were recorded for each lung (right and left) and three lung zones (upper, middle, and lower). They were recorded categorically for the amount detected, ranged as Absent, 1-25%, 26-50%, 51-75% and >75% for abnormality/lung fibrosis. For participants who received placebo/belumosudil in the DB period, the Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in the DB period. Number of participants with lung fibrosis at Baseline and Week 24 are reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: as for outcome 22
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 4 | 7 | 5
Participants
  Honeycombing Left Lung Zone 1 - Baseline: Absent: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Left Lung Zone 1 - Baseline: Absent | 4 | 7 | 4
  Honeycombing Left Lung Zone 1 - Baseline: 1-25%: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Left Lung Zone 1 - Baseline: 1-25% | 0 | 0 | 0
  Honeycombing Left Lung Zone 1 - Baseline: 26-50%: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Left Lung Zone 1 - Baseline: 26-50% | 0 | 0 | 0
  Honeycombing Left Lung Zone 1 - Baseline: 51-75%: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Left Lung Zone 1 - Baseline: 51-75% | 0 | 0 | 0
  Honeycombing Left Lung Zone 1 - Baseline: >75%: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Left Lung Zone 1 - Baseline: >75% | 0 | 0 | 0
  Honeycombing Left Lung Zone 1 - Week 24: Absent: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Left Lung Zone 1 - Week 24: Absent | 3 | 6 | 4
  Honeycombing Left Lung Zone 1 - Week 24: 1-25%: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Left Lung Zone 1 - Week 24: 1-25% | 1 | 0 | 1
  Honeycombing Left Lung Zone 1 - Week 24: 26-50%: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Left Lung Zone 1 - Week 24: 26-50% | 0 | 0 | 0
  Honeycombing Left Lung Zone 1 - Week 24: 51-75%: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Left Lung Zone 1 - Week 24: 51-75% | 0 | 0 | 0
  Honeycombing Left Lung Zone 1 - Week 24: >75%: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Left Lung Zone 1 - Week 24: >75% | 0 | 0 | 0
  Honeycombing Left Lung Zone 2 - Baseline: Absent: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Left Lung Zone 2 - Baseline: Absent | 4 | 7 | 4
  Honeycombing Left Lung Zone 2 - Baseline: 1-25%: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Left Lung Zone 2 - Baseline: 1-25% | 0 | 0 | 0
  Honeycombing Left Lung Zone 2 - Baseline: 26-50%: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Left Lung Zone 2 - Baseline: 26-50% | 0 | 0 | 0
  Honeycombing Left Lung Zone 2 - Baseline: 51-75%: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Left Lung Zone 2 - Baseline: 51-75% | 0 | 0 | 0
  Honeycombing Left Lung Zone 2 - Baseline: >75%: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Left Lung Zone 2 - Baseline: >75% | 0 | 0 | 0
  Honeycombing Left Lung Zone 2 - Week 24: Absent: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Left Lung Zone 2 - Week 24: Absent | 4 | 6 | 5
  Honeycombing Left Lung Zone 2 - Week 24: 1-25%: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Left Lung Zone 2 - Week 24: 1-25% | 0 | 0 | 0
  Honeycombing Left Lung Zone 2 - Week 24: 26-50%: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Left Lung Zone 2 - Week 24: 26-50% | 0 | 0 | 0
  Honeycombing Left Lung Zone 2 - Week 24: 51-75%: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Left Lung Zone 2 - Week 24: 51-75% | 0 | 0 | 0
  Honeycombing Left Lung Zone 2 - Week 24: >75%: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Left Lung Zone 2 - Week 24: >75% | 0 | 0 | 0
  Honeycombing Left Lung Zone 3 - Baseline: Absent: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Left Lung Zone 3 - Baseline: Absent | 4 | 5 | 4
  Honeycombing Left Lung Zone 3 - Baseline: 1-25%: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Left Lung Zone 3 - Baseline: 1-25% | 0 | 1 | 0
  Honeycombing Left Lung Zone 3 - Baseline: 26-50%: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Left Lung Zone 3 - Baseline: 26-50% | 0 | 1 | 0
  Honeycombing Left Lung Zone 3 - Baseline: 51-75%: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Left Lung Zone 3 - Baseline: 51-75% | 0 | 0 | 0
  Honeycombing Left Lung Zone 3 - Baseline: >75%: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Left Lung Zone 3 - Baseline: >75% | 0 | 0 | 0
  Honeycombing Left Lung Zone 3 - Week 24: Absent: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Left Lung Zone 3 - Week 24: Absent | 4 | 5 | 5
  Honeycombing Left Lung Zone 3 - Week 24: 1-25%: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Left Lung Zone 3 - Week 24: 1-25% | 0 | 1 | 0
  Honeycombing Left Lung Zone 3 - Week 24: 26-50%: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Left Lung Zone 3 - Week 24: 26-50% | 0 | 0 | 0
  Honeycombing Left Lung Zone 3 - Week 24: 51-75%: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Left Lung Zone 3 - Week 24: 51-75% | 0 | 0 | 0
  Honeycombing Left Lung Zone 3 - Week 24: >75%: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Left Lung Zone 3 - Week 24: >75% | 0 | 0 | 0
  Honeycombing Right Lung Zone 1 - Baseline: Absent: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Right Lung Zone 1 - Baseline: Absent | 4 | 7 | 4
  Honeycombing Right Lung Zone 1 - Baseline: 1-25%: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Right Lung Zone 1 - Baseline: 1-25% | 0 | 0 | 0
  Honeycombing Right Lung Zone 1 - Baseline: 26-50%: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Right Lung Zone 1 - Baseline: 26-50% | 0 | 0 | 0
  Honeycombing Right Lung Zone 1 - Baseline: 51-75%: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Right Lung Zone 1 - Baseline: 51-75% | 0 | 0 | 0
  Honeycombing Right Lung Zone 1 - Baseline: >75%: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Right Lung Zone 1 - Baseline: >75% | 0 | 0 | 0
  Honeycombing Right Lung Zone 1 - Week 24: Absent: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Right Lung Zone 1 - Week 24: Absent | 4 | 6 | 5
  Honeycombing Right Lung Zone 1 - Week 24: 1-25%: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Right Lung Zone 1 - Week 24: 1-25% | 0 | 0 | 0
  Honeycombing Right Lung Zone 1 - Week 24: 26-50%: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Right Lung Zone 1 - Week 24: 26-50% | 0 | 0 | 0
  Honeycombing Right Lung Zone 1 - Week 24: 51-75%: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Right Lung Zone 1 - Week 24: 51-75% | 0 | 0 | 0
  Honeycombing Right Lung Zone 1 - Week 24: >75%: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Right Lung Zone 1 - Week 24: >75% | 0 | 0 | 0
  Honeycombing Right Lung Zone 2 - Baseline: Absent: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Right Lung Zone 2 - Baseline: Absent | 4 | 7 | 4
  Honeycombing Right Lung Zone 2 - Baseline: 1-25%: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Right Lung Zone 2 - Baseline: 1-25% | 0 | 0 | 0
  Honeycombing Right Lung Zone 2 - Baseline: 26-50%: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Right Lung Zone 2 - Baseline: 26-50% | 0 | 0 | 0
  Honeycombing Right Lung Zone 2 - Baseline: 51-75%: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Right Lung Zone 2 - Baseline: 51-75% | 0 | 0 | 0
  Honeycombing Right Lung Zone 2 - Baseline: >75%: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Right Lung Zone 2 - Baseline: >75% | 0 | 0 | 0
  Honeycombing Right Lung Zone 2 - Week 24: Absent: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Right Lung Zone 2 - Week 24: Absent | 4 | 6 | 5
  Honeycombing Right Lung Zone 2 - Week 24: 1-25%: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Right Lung Zone 2 - Week 24: 1-25% | 0 | 0 | 0
  Honeycombing Right Lung Zone 2 - Week 24: 26-50%: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Right Lung Zone 2 - Week 24: 26-50% | 0 | 0 | 0
  Honeycombing Right Lung Zone 2 - Week 24: 51-75%: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Right Lung Zone 2 - Week 24: 51-75% | 0 | 0 | 0
  Honeycombing Right Lung Zone 2 - Week 24: >75%: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Right Lung Zone 2 - Week 24: >75% | 0 | 0 | 0
  Honeycombing Right Lung Zone 3 - Baseline: Absent: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Right Lung Zone 3 - Baseline: Absent | 4 | 5 | 4
  Honeycombing Right Lung Zone 3 - Baseline: 1-25%: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Right Lung Zone 3 - Baseline: 1-25% | 0 | 1 | 0
  Honeycombing Right Lung Zone 3 - Baseline: 26-50%: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Right Lung Zone 3 - Baseline: 26-50% | 0 | 1 | 0
  Honeycombing Right Lung Zone 3 - Baseline: 51-75%: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Right Lung Zone 3 - Baseline: 51-75% | 0 | 0 | 0
  Honeycombing Right Lung Zone 3 - Baseline: >75%: number analyzed (Participants) | 4 | 7 | 4
  Honeycombing Right Lung Zone 3 - Baseline: >75% | 0 | 0 | 0
  Honeycombing Right Lung Zone 3 - Week 24: Absent: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Right Lung Zone 3 - Week 24: Absent | 4 | 5 | 5
  Honeycombing Right Lung Zone 3 - Week 24: 1-25%: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Right Lung Zone 3 - Week 24: 1-25% | 0 | 1 | 0
  Honeycombing Right Lung Zone 3 - Week 24: 26-50%: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Right Lung Zone 3 - Week 24: 26-50% | 0 | 0 | 0
  Honeycombing Right Lung Zone 3 - Week 24: 51-75%: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Right Lung Zone 3 - Week 24: 51-75% | 0 | 0 | 0
  Honeycombing Right Lung Zone 3 - Week 24: >75%: number analyzed (Participants) | 4 | 6 | 5
  Honeycombing Right Lung Zone 3 - Week 24: >75% | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 1 - Baseline: Absent: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Left Lung Zone 1 - Baseline: Absent | 3 | 6 | 4
  Pulmonary Fibrosis Left Lung Zone 1 - Baseline: 1-25%: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Left Lung Zone 1 - Baseline: 1-25% | 1 | 1 | 0
  Pulmonary Fibrosis Left Lung Zone 1 - Baseline: 26-50%: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Left Lung Zone 1 - Baseline: 26-50% | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 1 - Baseline: 51-75%: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Left Lung Zone 1 - Baseline: 51-75% | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 1 - Baseline: >75%: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Left Lung Zone 1 - Baseline: >75% | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 1 - Week 24: Absent: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Left Lung Zone 1 - Week 24: Absent | 3 | 6 | 5
  Pulmonary Fibrosis Left Lung Zone 1 - Week 24: 1-25%: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Left Lung Zone 1 - Week 24: 1-25% | 1 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 1 - Week 24: 26-50%: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Left Lung Zone 1 - Week 24: 26-50% | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 1 - Week 24: 51-75%: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Left Lung Zone 1 - Week 24: 51-75% | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 1 - Week 24: >75%: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Left Lung Zone 1 - Week 24: >75% | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 2 - Baseline: Absent: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Left Lung Zone 2 - Baseline: Absent | 4 | 4 | 4
  Pulmonary Fibrosis Left Lung Zone 2 - Baseline: 1-25%: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Left Lung Zone 2 - Baseline: 1-25% | 0 | 3 | 0
  Pulmonary Fibrosis Left Lung Zone 2 - Baseline: 26-50%: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Left Lung Zone 2 - Baseline: 26-50% | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 2 - Baseline: 51-75%: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Left Lung Zone 2 - Baseline: 51-75% | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 2 - Baseline: >75%: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Left Lung Zone 2 - Baseline: >75% | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 2 - Week 24: Absent: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Left Lung Zone 2 - Week 24: Absent | 4 | 3 | 4
  Pulmonary Fibrosis Left Lung Zone 2 - Week 24: 1-25%: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Left Lung Zone 2 - Week 24: 1-25% | 0 | 3 | 1
  Pulmonary Fibrosis Left Lung Zone 2 - Week 24: 26-50%: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Left Lung Zone 2 - Week 24: 26-50% | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 2 - Week 24: 51-75%: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Left Lung Zone 2 - Week 24: 51-75% | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 2 - Week 24: >75%: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Left Lung Zone 2 - Week 24: >75% | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 3 - Baseline: Absent: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Left Lung Zone 3 - Baseline: Absent | 4 | 1 | 2
  Pulmonary Fibrosis Left Lung Zone 3 - Baseline: 1-25%: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Left Lung Zone 3 - Baseline: 1-25% | 0 | 2 | 1
  Pulmonary Fibrosis Left Lung Zone 3 - Baseline: 26-50%: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Left Lung Zone 3 - Baseline: 26-50% | 0 | 2 | 1
  Pulmonary Fibrosis Left Lung Zone 3 - Baseline: 51-75%: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Left Lung Zone 3 - Baseline: 51-75% | 0 | 1 | 0
  Pulmonary Fibrosis Left Lung Zone 3 - Baseline: >75%: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Left Lung Zone 3 - Baseline: >75% | 0 | 1 | 0
  Pulmonary Fibrosis Left Lung Zone 3 - Week 24: Absent: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Left Lung Zone 3 - Week 24: Absent | 2 | 1 | 0
  Pulmonary Fibrosis Left Lung Zone 3 - Week 24: 1-25%: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Left Lung Zone 3 - Week 24: 1-25% | 2 | 3 | 4
  Pulmonary Fibrosis Left Lung Zone 3 - Week 24: 26-50%: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Left Lung Zone 3 - Week 24: 26-50% | 0 | 1 | 1
  Pulmonary Fibrosis Left Lung Zone 3 - Week 24: 51-75%: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Left Lung Zone 3 - Week 24: 51-75% | 0 | 1 | 0
  Pulmonary Fibrosis Left Lung Zone 3 - Week 24: >75%: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Left Lung Zone 3 - Week 24: >75% | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 1 - Baseline: Absent: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Right Lung Zone 1 - Baseline: Absent | 4 | 6 | 4
  Pulmonary Fibrosis Right Lung Zone 1 - Baseline: 1-25%: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Right Lung Zone 1 - Baseline: 1-25% | 0 | 1 | 0
  Pulmonary Fibrosis Right Lung Zone 1 - Baseline: 26-50%: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Right Lung Zone 1 - Baseline: 26-50% | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 1 - Baseline: 51-75%: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Right Lung Zone 1 - Baseline: 51-75% | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 1 - Baseline: >75%: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Right Lung Zone 1 - Baseline: >75% | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 1 - Week 24: Absent: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Right Lung Zone 1 - Week 24: Absent | 2 | 5 | 3
  Pulmonary Fibrosis Right Lung Zone 1 - Week 24: 1-25%: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Right Lung Zone 1 - Week 24: 1-25% | 2 | 1 | 2
  Pulmonary Fibrosis Right Lung Zone 1 - Week 24: 26-50%: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Right Lung Zone 1 - Week 24: 26-50% | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 1 - Week 24: 51-75%: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Right Lung Zone 1 - Week 24: 51-75% | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 1 - Week 24: >75%: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Right Lung Zone 1 - Week 24: >75% | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 2 - Baseline: Absent: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Right Lung Zone 2 - Baseline: Absent | 4 | 3 | 3
  Pulmonary Fibrosis Right Lung Zone 2 - Baseline: 1-25%: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Right Lung Zone 2 - Baseline: 1-25% | 0 | 4 | 1
  Pulmonary Fibrosis Right Lung Zone 2 - Baseline: 26-50%: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Right Lung Zone 2 - Baseline: 26-50% | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 2 - Baseline: 51-75%: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Right Lung Zone 2 - Baseline: 51-75% | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 2 - Baseline: >75%: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Right Lung Zone 2 - Baseline: >75% | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 2 - Week 24: Absent: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Right Lung Zone 2 - Week 24: Absent | 4 | 4 | 3
  Pulmonary Fibrosis Right Lung Zone 2 - Week 24: 1-25%: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Right Lung Zone 2 - Week 24: 1-25% | 0 | 2 | 1
  Pulmonary Fibrosis Right Lung Zone 2 - Week 24: 26-50%: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Right Lung Zone 2 - Week 24: 26-50% | 0 | 0 | 1
  Pulmonary Fibrosis Right Lung Zone 2 - Week 24: 51-75%: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Right Lung Zone 2 - Week 24: 51-75% | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 2 - Week 24: >75%: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Right Lung Zone 2 - Week 24: >75% | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 3 - Baseline: Absent: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Right Lung Zone 3 - Baseline: Absent | 3 | 1 | 0
  Pulmonary Fibrosis Right Lung Zone 3 - Baseline: 1-25%: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Right Lung Zone 3 - Baseline: 1-25% | 1 | 2 | 2
  Pulmonary Fibrosis Right Lung Zone 3 - Baseline: 26-50%: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Right Lung Zone 3 - Baseline: 26-50% | 0 | 2 | 2
  Pulmonary Fibrosis Right Lung Zone 3 - Baseline: 51-75%: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Right Lung Zone 3 - Baseline: 51-75% | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 3 - Baseline: >75%: number analyzed (Participants) | 4 | 7 | 4
  Pulmonary Fibrosis Right Lung Zone 3 - Baseline: >75% | 0 | 2 | 0
  Pulmonary Fibrosis Right Lung Zone 3 - Week 24: Absent: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Right Lung Zone 3 - Week 24: Absent | 2 | 2 | 0
  Pulmonary Fibrosis Right Lung Zone 3 - Week 24: 1-25%: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Right Lung Zone 3 - Week 24: 1-25% | 2 | 2 | 3
  Pulmonary Fibrosis Right Lung Zone 3 - Week 24: 26-50%: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Right Lung Zone 3 - Week 24: 26-50% | 0 | 1 | 2
  Pulmonary Fibrosis Right Lung Zone 3 - Week 24: 51-75%: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Right Lung Zone 3 - Week 24: 51-75% | 0 | 1 | 0
  Pulmonary Fibrosis Right Lung Zone 3 - Week 24: >75%: number analyzed (Participants) | 4 | 6 | 5
  Pulmonary Fibrosis Right Lung Zone 3 - Week 24: >75% | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 1 - Baseline: Absent: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Left Lung Zone 1 - Baseline: Absent | 2 | 4 | 3
  Pure Ground-Glass Opacity Left Lung Zone 1 - Baseline: 1-25%: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Left Lung Zone 1 - Baseline: 1-25% | 2 | 3 | 1
  Pure Ground-Glass Opacity Left Lung Zone 1 - Baseline: 26-50%: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Left Lung Zone 1 - Baseline: 26-50% | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 1 - Baseline: 51-75%: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Left Lung Zone 1 - Baseline: 51-75% | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 1 - Baseline: >75%: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Left Lung Zone 1 - Baseline: >75% | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 1 - Week 24: Absent: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Left Lung Zone 1 - Week 24: Absent | 4 | 4 | 4
  Pure Ground-Glass Opacity Left Lung Zone 1 - Week 24: 1-25%: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Left Lung Zone 1 - Week 24: 1-25% | 0 | 2 | 1
  Pure Ground-Glass Opacity Left Lung Zone 1 - Week 24: 26-50%: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Left Lung Zone 1 - Week 24: 26-50% | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 1 - Week 24: 51-75%: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Left Lung Zone 1 - Week 24: 51-75% | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 1 - Week 24: >75%: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Left Lung Zone 1 - Week 24: >75% | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 2 - Baseline: Absent: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Left Lung Zone 2 - Baseline: Absent | 3 | 4 | 3
  Pure Ground-Glass Opacity Left Lung Zone 2 - Baseline: 1-25%: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Left Lung Zone 2 - Baseline: 1-25% | 1 | 3 | 1
  Pure Ground-Glass Opacity Left Lung Zone 2 - Baseline: 26-50%: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Left Lung Zone 2 - Baseline: 26-50% | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 2 - Baseline: 51-75%: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Left Lung Zone 2 - Baseline: 51-75% | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 2 - Baseline: >75%: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Left Lung Zone 2 - Baseline: >75% | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 2 - Week 24: Absent: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Left Lung Zone 2 - Week 24: Absent | 4 | 3 | 4
  Pure Ground-Glass Opacity Left Lung Zone 2 - Week 24: 1-25%: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Left Lung Zone 2 - Week 24: 1-25% | 0 | 3 | 1
  Pure Ground-Glass Opacity Left Lung Zone 2 - Week 24: 26-50%: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Left Lung Zone 2 - Week 24: 26-50% | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 2 - Week 24: 51-75%: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Left Lung Zone 2 - Week 24: 51-75% | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 2 - Week 24: >75%: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Left Lung Zone 2 - Week 24: >75% | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 3 - Baseline: Absent: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Left Lung Zone 3 - Baseline: Absent | 2 | 4 | 2
  Pure Ground-Glass Opacity Left Lung Zone 3 - Baseline: 1-25%: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Left Lung Zone 3 - Baseline: 1-25% | 1 | 3 | 2
  Pure Ground-Glass Opacity Left Lung Zone 3 - Baseline: 26-50%: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Left Lung Zone 3 - Baseline: 26-50% | 1 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 3 - Baseline: 51-75%: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Left Lung Zone 3 - Baseline: 51-75% | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 3 - Baseline: >75%: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Left Lung Zone 3 - Baseline: >75% | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 3 - Week 24: Absent: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Left Lung Zone 3 - Week 24: Absent | 2 | 2 | 2
  Pure Ground-Glass Opacity Left Lung Zone 3 - Week 24: 1-25%: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Left Lung Zone 3 - Week 24: 1-25% | 2 | 2 | 2
  Pure Ground-Glass Opacity Left Lung Zone 3 - Week 24: 26-50%: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Left Lung Zone 3 - Week 24: 26-50% | 0 | 1 | 1
  Pure Ground-Glass Opacity Left Lung Zone 3 - Week 24: 51-75%: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Left Lung Zone 3 - Week 24: 51-75% | 0 | 1 | 0
  Pure Ground-Glass Opacity Left Lung Zone 3 - Week 24: >75%: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Left Lung Zone 3 - Week 24: >75% | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 1 - Baseline: Absent: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Right Lung Zone 1 - Baseline: Absent | 3 | 4 | 2
  Pure Ground-Glass Opacity Right Lung Zone 1 - Baseline: 1-25%: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Right Lung Zone 1 - Baseline: 1-25% | 1 | 2 | 2
  Pure Ground-Glass Opacity Right Lung Zone 1 - Baseline: 26-50%: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Right Lung Zone 1 - Baseline: 26-50% | 0 | 1 | 0
  Pure Ground-Glass Opacity Right Lung Zone 1 - Baseline: 51-75%: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Right Lung Zone 1 - Baseline: 51-75% | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 1 - Baseline: >75%: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Right Lung Zone 1 - Baseline: >75% | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 1 - Week 24: Absent: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Right Lung Zone 1 - Week 24: Absent | 3 | 3 | 3
  Pure Ground-Glass Opacity Right Lung Zone 1 - Week 24: 1-25%: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Right Lung Zone 1 - Week 24: 1-25% | 1 | 2 | 2
  Pure Ground-Glass Opacity Right Lung Zone 1 - Week 24: 26-50%: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Right Lung Zone 1 - Week 24: 26-50% | 0 | 1 | 0
  Pure Ground-Glass Opacity Right Lung Zone 1 - Week 24: 51-75%: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Right Lung Zone 1 - Week 24: 51-75% | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 1 - Week 24: >75%: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Right Lung Zone 1 - Week 24: >75% | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 2 - Baseline: Absent: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Right Lung Zone 2 - Baseline: Absent | 3 | 5 | 2
  Pure Ground-Glass Opacity Right Lung Zone 2 - Baseline: 1-25%: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Right Lung Zone 2 - Baseline: 1-25% | 1 | 1 | 2
  Pure Ground-Glass Opacity Right Lung Zone 2 - Baseline: 26-50%: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Right Lung Zone 2 - Baseline: 26-50% | 0 | 1 | 0
  Pure Ground-Glass Opacity Right Lung Zone 2 - Baseline: 51-75%: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Right Lung Zone 2 - Baseline: 51-75% | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 2 - Baseline: >75%: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Right Lung Zone 2 - Baseline: >75% | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 2 - Week 24: Absent: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Right Lung Zone 2 - Week 24: Absent | 3 | 4 | 3
  Pure Ground-Glass Opacity Right Lung Zone 2 - Week 24: 1-25%: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Right Lung Zone 2 - Week 24: 1-25% | 1 | 2 | 2
  Pure Ground-Glass Opacity Right Lung Zone 2 - Week 24: 26-50%: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Right Lung Zone 2 - Week 24: 26-50% | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 2 - Week 24: 51-75%: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Right Lung Zone 2 - Week 24: 51-75% | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 2 - Week 24: >75%: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Right Lung Zone 2 - Week 24: >75% | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 3 - Baseline: Absent: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Right Lung Zone 3 - Baseline: Absent | 2 | 3 | 1
  Pure Ground-Glass Opacity Right Lung Zone 3 - Baseline: 1-25%: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Right Lung Zone 3 - Baseline: 1-25% | 1 | 3 | 3
  Pure Ground-Glass Opacity Right Lung Zone 3 - Baseline: 26-50%: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Right Lung Zone 3 - Baseline: 26-50% | 1 | 1 | 0
  Pure Ground-Glass Opacity Right Lung Zone 3 - Baseline: 51-75%: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Right Lung Zone 3 - Baseline: 51-75% | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 3 - Baseline: >75%: number analyzed (Participants) | 4 | 7 | 4
  Pure Ground-Glass Opacity Right Lung Zone 3 - Baseline: >75% | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 3 - Week 24: Absent: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Right Lung Zone 3 - Week 24: Absent | 2 | 2 | 1
  Pure Ground-Glass Opacity Right Lung Zone 3 - Week 24: 1-25%: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Right Lung Zone 3 - Week 24: 1-25% | 2 | 3 | 4
  Pure Ground-Glass Opacity Right Lung Zone 3 - Week 24: 26-50%: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Right Lung Zone 3 - Week 24: 26-50% | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 3 - Week 24: 51-75%: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Right Lung Zone 3 - Week 24: 51-75% | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 3 - Week 24: >75%: number analyzed (Participants) | 4 | 6 | 5
  Pure Ground-Glass Opacity Right Lung Zone 3 - Week 24: >75% | 0 | 1 | 0

33. Secondary Outcome: OLE Period: Number of Participants With Lung Fibrosis at Baseline and Week 52-ILD Participants
Description: Lung fibrosis is a lung disease in which lung tissue becomes damaged and scared. Lung fibrosis was assessed using HRCT. HRCT is a type of computed tomography used to diagnose and stage the severity. Pure ground-class opacity, pulmonary fibrosis and honeycombing were recorded for each lung (right and left) and three lung zones (upper, middle, and lower). They were recorded categorically for the amount detected, ranged as Absent, 1-25%, 26-50%, 51-75% and >75% for abnormality/lung fibrosis. Number of participants with lung fibrosis at Baseline and Week 52 are reported in this outcome measure. In the data table below, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Time Frame: Baseline, Week 52
Population: Analysis was performed on participants with ILD. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline: valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value: valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period.
Measure: Count of Participants; unit: Participants
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 4 | 2 | 6 | 3
Participants
  Honeycombing Left Lung Zone 1 - Baseline: Absent | 4 | 2 | 6 | 2
  Honeycombing Left Lung Zone 1 - Baseline: 1-25% | 0 | 0 | 0 | 1
  Honeycombing Left Lung Zone 1 - Baseline: 26-50% | 0 | 0 | 0 | 0
  Honeycombing Left Lung Zone 1 - Baseline: 51-75% | 0 | 0 | 0 | 0
  Honeycombing Left Lung Zone 1 - Baseline: >75% | 0 | 0 | 0 | 0
  Honeycombing Left Lung Zone 1 - Week 52: Absent: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Left Lung Zone 1 - Week 52: Absent | 4 | 2 | 3 | 3
  Honeycombing Left Lung Zone 1 - Week 52: 1-25%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Left Lung Zone 1 - Week 52: 1-25% | 0 | 0 | 0 | 0
  Honeycombing Left Lung Zone 1 - Week 52: 26-50%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Left Lung Zone 1 - Week 52: 26-50% | 0 | 0 | 0 | 0
  Honeycombing Left Lung Zone 1 - Week 52: 51-75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Left Lung Zone 1 - Week 52: 51-75% | 0 | 0 | 0 | 0
  Honeycombing Left Lung Zone 1 - Week 52: >75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Left Lung Zone 1 - Week 52: >75% | 0 | 0 | 0 | 0
  Honeycombing Left Lung Zone 2 - Baseline: Absent | 4 | 2 | 6 | 3
  Honeycombing Left Lung Zone 2 - Baseline: 1-25% | 0 | 0 | 0 | 0
  Honeycombing Left Lung Zone 2 - Baseline: 26-50% | 0 | 0 | 0 | 0
  Honeycombing Left Lung Zone 2 - Baseline: 51-75% | 0 | 0 | 0 | 0
  Honeycombing Left Lung Zone 2 - Baseline: >75% | 0 | 0 | 0 | 0
  Honeycombing Left Lung Zone 2 - Week 52: Absent: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Left Lung Zone 2 - Week 52: Absent | 4 | 2 | 3 | 3
  Honeycombing Left Lung Zone 2 - Week 52: 1-25%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Left Lung Zone 2 - Week 52: 1-25% | 0 | 0 | 0 | 0
  Honeycombing Left Lung Zone 2 - Week 52: 26-50%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Left Lung Zone 2 - Week 52: 26-50% | 0 | 0 | 0 | 0
  Honeycombing Left Lung Zone 2 - Week 52: 51-75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Left Lung Zone 2 - Week 52: 51-75% | 0 | 0 | 0 | 0
  Honeycombing Left Lung Zone 2 - Week 52: >75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Left Lung Zone 2 - Week 52: >75% | 0 | 0 | 0 | 0
  Honeycombing Left Lung Zone 3 - Baseline: Absent | 4 | 2 | 5 | 3
  Honeycombing Left Lung Zone 3 - Baseline: 1-25% | 0 | 0 | 0 | 0
  Honeycombing Left Lung Zone 3 - Baseline: 26-50% | 0 | 0 | 1 | 0
  Honeycombing Left Lung Zone 3 - Baseline: 51-75% | 0 | 0 | 0 | 0
  Honeycombing Left Lung Zone 3 - Baseline: >75% | 0 | 0 | 0 | 0
  Honeycombing Left Lung Zone 3 - Week 52: Absent: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Left Lung Zone 3 - Week 52: Absent | 4 | 2 | 2 | 3
  Honeycombing Left Lung Zone 3 - Week 52: 1-25%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Left Lung Zone 3 - Week 52: 1-25% | 0 | 0 | 1 | 0
  Honeycombing Left Lung Zone 3 - Week 52: 26-50%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Left Lung Zone 3 - Week 52: 26-50% | 0 | 0 | 0 | 0
  Honeycombing Left Lung Zone 3 - Week 52: 51-75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Left Lung Zone 3 - Week 52: 51-75% | 0 | 0 | 0 | 0
  Honeycombing Left Lung Zone 3 - Week 52: >75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Left Lung Zone 3 - Week 52: >75% | 0 | 0 | 0 | 0
  Honeycombing Right Lung Zone 1 - Baseline: Absent | 4 | 2 | 6 | 3
  Honeycombing Right Lung Zone 1 - Baseline: 1-25% | 0 | 0 | 0 | 0
  Honeycombing Right Lung Zone 1 - Baseline: 26-50% | 0 | 0 | 0 | 0
  Honeycombing Right Lung Zone 1 - Baseline: 51-75% | 0 | 0 | 0 | 0
  Honeycombing Right Lung Zone 1 - Baseline: >75% | 0 | 0 | 0 | 0
  Honeycombing Right Lung Zone 1 - Week 52: Absent: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Right Lung Zone 1 - Week 52: Absent | 4 | 2 | 3 | 3
  Honeycombing Right Lung Zone 1 - Week 52: 1-25%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Right Lung Zone 1 - Week 52: 1-25% | 0 | 0 | 0 | 0
  Honeycombing Right Lung Zone 1 - Week 52: 26-50%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Right Lung Zone 1 - Week 52: 26-50% | 0 | 0 | 0 | 0
  Honeycombing Right Lung Zone 1 - Week 52: 51-75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Right Lung Zone 1 - Week 52: 51-75% | 0 | 0 | 0 | 0
  Honeycombing Right Lung Zone 1 - Week 52: >75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Right Lung Zone 1 - Week 52: >75% | 0 | 0 | 0 | 0
  Honeycombing Right Lung Zone 2 - Baseline: Absent | 4 | 2 | 6 | 3
  Honeycombing Right Lung Zone 2 - Baseline: 1-25% | 0 | 0 | 0 | 0
  Honeycombing Right Lung Zone 2 - Baseline: 26-50% | 0 | 0 | 0 | 0
  Honeycombing Right Lung Zone 2 - Baseline: 51-75% | 0 | 0 | 0 | 0
  Honeycombing Right Lung Zone 2 - Baseline: >75% | 0 | 0 | 0 | 0
  Honeycombing Right Lung Zone 2 - Week 52: Absent: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Right Lung Zone 2 - Week 52: Absent | 4 | 2 | 3 | 3
  Honeycombing Right Lung Zone 2 - Week 52: 1-25%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Right Lung Zone 2 - Week 52: 1-25% | 0 | 0 | 0 | 0
  Honeycombing Right Lung Zone 2 - Week 52: 26-50%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Right Lung Zone 2 - Week 52: 26-50% | 0 | 0 | 0 | 0
  Honeycombing Right Lung Zone 2 - Week 52: 51-75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Right Lung Zone 2 - Week 52: 51-75% | 0 | 0 | 0 | 0
  Honeycombing Right Lung Zone 2 - Week 52: >75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Right Lung Zone 2 - Week 52: >75% | 0 | 0 | 0 | 0
  Honeycombing Right Lung Zone 3 - Baseline: Absent | 4 | 2 | 5 | 3
  Honeycombing Right Lung Zone 3 - Baseline: 1-25% | 0 | 0 | 0 | 0
  Honeycombing Right Lung Zone 3 - Baseline: 26-50% | 0 | 0 | 1 | 0
  Honeycombing Right Lung Zone 3 - Baseline: 51-75% | 0 | 0 | 0 | 0
  Honeycombing Right Lung Zone 3 - Baseline: >75% | 0 | 0 | 0 | 0
  Honeycombing Right Lung Zone 3 - Week 52: Absent: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Right Lung Zone 3 - Week 52: Absent | 4 | 2 | 3 | 3
  Honeycombing Right Lung Zone 3 - Week 52: 1-25%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Right Lung Zone 3 - Week 52: 1-25% | 0 | 0 | 0 | 0
  Honeycombing Right Lung Zone 3 - Week 52: 26-50%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Right Lung Zone 3 - Week 52: 26-50% | 0 | 0 | 0 | 0
  Honeycombing Right Lung Zone 3 - Week 52: 51-75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Right Lung Zone 3 - Week 52: 51-75% | 0 | 0 | 0 | 0
  Honeycombing Right Lung Zone 3 - Week 52: >75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Honeycombing Right Lung Zone 3 - Week 52: >75% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 1 - Baseline: Absent | 3 | 2 | 6 | 3
  Pulmonary Fibrosis Left Lung Zone 1 - Baseline: 1-25% | 1 | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 1 - Baseline: 26-50% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 1 - Baseline: 51-75% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 1 - Baseline: >75% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 1 - Week 52: Absent: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Left Lung Zone 1 - Week 52: Absent | 3 | 2 | 2 | 1
  Pulmonary Fibrosis Left Lung Zone 1 - Week 52: 1-25%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Left Lung Zone 1 - Week 52: 1-25% | 1 | 0 | 1 | 2
  Pulmonary Fibrosis Left Lung Zone 1 - Week 52: 26-50%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Left Lung Zone 1 - Week 52: 26-50% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 1 - Week 52: 51-75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Left Lung Zone 1 - Week 52: 51-75% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 1 - Week 52: >75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Left Lung Zone 1 - Week 52: >75% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 2 - Baseline: Absent | 4 | 2 | 4 | 2
  Pulmonary Fibrosis Left Lung Zone 2 - Baseline: 1-25% | 0 | 0 | 2 | 1
  Pulmonary Fibrosis Left Lung Zone 2 - Baseline: 26-50% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 2 - Baseline: 51-75% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 2 - Baseline: >75% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 2 - Week 52: Absent: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Left Lung Zone 2 - Week 52: Absent | 4 | 1 | 3 | 3
  Pulmonary Fibrosis Left Lung Zone 2 - Week 52: 1-25%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Left Lung Zone 2 - Week 52: 1-25% | 0 | 1 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 2 - Week 52: 26-50%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Left Lung Zone 2 - Week 52: 26-50% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 2 - Week 52: 51-75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Left Lung Zone 2 - Week 52: 51-75% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 2 - Week 52: >75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Left Lung Zone 2 - Week 52: >75% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 3 - Baseline: Absent | 4 | 0 | 1 | 0
  Pulmonary Fibrosis Left Lung Zone 3 - Baseline: 1-25% | 0 | 2 | 2 | 2
  Pulmonary Fibrosis Left Lung Zone 3 - Baseline: 26-50% | 0 | 0 | 2 | 1
  Pulmonary Fibrosis Left Lung Zone 3 - Baseline: 51-75% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Left Lung Zone 3 - Baseline: >75% | 0 | 0 | 1 | 0
  Pulmonary Fibrosis Left Lung Zone 3 - Week 52: Absent: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Left Lung Zone 3 - Week 52: Absent | 3 | 0 | 1 | 1
  Pulmonary Fibrosis Left Lung Zone 3 - Week 52: 1-25%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Left Lung Zone 3 - Week 52: 1-25% | 1 | 1 | 1 | 0
  Pulmonary Fibrosis Left Lung Zone 3 - Week 52: 26-50%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Left Lung Zone 3 - Week 52: 26-50% | 0 | 1 | 0 | 2
  Pulmonary Fibrosis Left Lung Zone 3 - Week 52: 51-75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Left Lung Zone 3 - Week 52: 51-75% | 0 | 0 | 1 | 0
  Pulmonary Fibrosis Left Lung Zone 3 - Week 52: >75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Left Lung Zone 3 - Week 52: >75% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 1 - Baseline: Absent | 4 | 2 | 6 | 1
  Pulmonary Fibrosis Right Lung Zone 1 - Baseline: 1-25% | 0 | 0 | 0 | 2
  Pulmonary Fibrosis Right Lung Zone 1 - Baseline: 26-50% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 1 - Baseline: 51-75% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 1 - Baseline: >75% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 1 - Week 52: Absent: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Right Lung Zone 1 - Week 52: Absent | 3 | 2 | 2 | 1
  Pulmonary Fibrosis Right Lung Zone 1 - Week 52: 1-25%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Right Lung Zone 1 - Week 52: 1-25% | 1 | 0 | 1 | 2
  Pulmonary Fibrosis Right Lung Zone 1 - Week 52: 26-50%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Right Lung Zone 1 - Week 52: 26-50% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 1 - Week 52: 51-75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Right Lung Zone 1 - Week 52: 51-75% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 1 - Week 52: >75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Right Lung Zone 1 - Week 52: >75% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 2 - Baseline: Absent | 4 | 2 | 3 | 1
  Pulmonary Fibrosis Right Lung Zone 2 - Baseline: 1-25% | 0 | 0 | 3 | 1
  Pulmonary Fibrosis Right Lung Zone 2 - Baseline: 26-50% | 0 | 0 | 0 | 1
  Pulmonary Fibrosis Right Lung Zone 2 - Baseline: 51-75% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 2 - Baseline: >75% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 2 - Week 52: Absent: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Right Lung Zone 2 - Week 52: Absent | 3 | 1 | 1 | 0
  Pulmonary Fibrosis Right Lung Zone 2 - Week 52: 1-25%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Right Lung Zone 2 - Week 52: 1-25% | 1 | 1 | 2 | 2
  Pulmonary Fibrosis Right Lung Zone 2 - Week 52: 26-50%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Right Lung Zone 2 - Week 52: 26-50% | 0 | 0 | 0 | 1
  Pulmonary Fibrosis Right Lung Zone 2 - Week 52: 51-75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Right Lung Zone 2 - Week 52: 51-75% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 2 - Week 52: >75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Right Lung Zone 2 - Week 52: >75% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 3 - Baseline: Absent | 3 | 0 | 1 | 0
  Pulmonary Fibrosis Right Lung Zone 3 - Baseline: 1-25% | 1 | 2 | 2 | 1
  Pulmonary Fibrosis Right Lung Zone 3 - Baseline: 26-50% | 0 | 0 | 2 | 2
  Pulmonary Fibrosis Right Lung Zone 3 - Baseline: 51-75% | 0 | 0 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 3 - Baseline: >75% | 0 | 0 | 1 | 0
  Pulmonary Fibrosis Right Lung Zone 3 - Week 52: Absent: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Right Lung Zone 3 - Week 52: Absent | 2 | 0 | 1 | 1
  Pulmonary Fibrosis Right Lung Zone 3 - Week 52: 1-25%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Right Lung Zone 3 - Week 52: 1-25% | 2 | 1 | 1 | 0
  Pulmonary Fibrosis Right Lung Zone 3 - Week 52: 26-50%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Right Lung Zone 3 - Week 52: 26-50% | 0 | 0 | 1 | 2
  Pulmonary Fibrosis Right Lung Zone 3 - Week 52: 51-75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Right Lung Zone 3 - Week 52: 51-75% | 0 | 1 | 0 | 0
  Pulmonary Fibrosis Right Lung Zone 3 - Week 52: >75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pulmonary Fibrosis Right Lung Zone 3 - Week 52: >75% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 1 - Baseline: Absent | 2 | 2 | 3 | 2
  Pure Ground-Glass Opacity Left Lung Zone 1 - Baseline: 1-25% | 2 | 0 | 3 | 1
  Pure Ground-Glass Opacity Left Lung Zone 1 - Baseline: 26-50% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 1 - Baseline: 51-75% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 1 - Baseline: >75% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 1 - Week 52: Absent: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Left Lung Zone 1 - Week 52: Absent | 4 | 1 | 3 | 2
  Pure Ground-Glass Opacity Left Lung Zone 1 - Week 52: 1-25%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Left Lung Zone 1 - Week 52: 1-25% | 0 | 1 | 0 | 1
  Pure Ground-Glass Opacity Left Lung Zone 1 - Week 52: 26-50%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Left Lung Zone 1 - Week 52: 26-50% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 1 - Week 52: 51-75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Left Lung Zone 1 - Week 52: 51-75% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 1 - Week 52: >75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Left Lung Zone 1 - Week 52: >75% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 2 - Baseline: Absent | 3 | 2 | 4 | 2
  Pure Ground-Glass Opacity Left Lung Zone 2 - Baseline: 1-25% | 1 | 0 | 2 | 1
  Pure Ground-Glass Opacity Left Lung Zone 2 - Baseline: 26-50% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 2 - Baseline: 51-75% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 2 - Baseline: >75% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 2 - Week 52: Absent: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Left Lung Zone 2 - Week 52: Absent | 4 | 2 | 2 | 2
  Pure Ground-Glass Opacity Left Lung Zone 2 - Week 52: 1-25%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Left Lung Zone 2 - Week 52: 1-25% | 0 | 0 | 0 | 1
  Pure Ground-Glass Opacity Left Lung Zone 2 - Week 52: 26-50%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Left Lung Zone 2 - Week 52: 26-50% | 0 | 0 | 1 | 0
  Pure Ground-Glass Opacity Left Lung Zone 2 - Week 52: 51-75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Left Lung Zone 2 - Week 52: 51-75% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 2 - Week 52: >75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Left Lung Zone 2 - Week 52: >75% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 3 - Baseline: Absent | 2 | 1 | 4 | 1
  Pure Ground-Glass Opacity Left Lung Zone 3 - Baseline: 1-25% | 1 | 1 | 2 | 1
  Pure Ground-Glass Opacity Left Lung Zone 3 - Baseline: 26-50% | 1 | 0 | 0 | 1
  Pure Ground-Glass Opacity Left Lung Zone 3 - Baseline: 51-75% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 3 - Baseline: >75% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 3 - Week 52: Absent: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Left Lung Zone 3 - Week 52: Absent | 1 | 1 | 1 | 0
  Pure Ground-Glass Opacity Left Lung Zone 3 - Week 52: 1-25%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Left Lung Zone 3 - Week 52: 1-25% | 2 | 1 | 2 | 3
  Pure Ground-Glass Opacity Left Lung Zone 3 - Week 52: 26-50%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Left Lung Zone 3 - Week 52: 26-50% | 1 | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 3 - Week 52: 51-75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Left Lung Zone 3 - Week 52: 51-75% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Left Lung Zone 3 - Week 52: >75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Left Lung Zone 3 - Week 52: >75% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 1 - Baseline: Absent | 3 | 1 | 3 | 2
  Pure Ground-Glass Opacity Right Lung Zone 1 - Baseline: 1-25% | 1 | 1 | 2 | 1
  Pure Ground-Glass Opacity Right Lung Zone 1 - Baseline: 26-50% | 0 | 0 | 1 | 0
  Pure Ground-Glass Opacity Right Lung Zone 1 - Baseline: 51-75% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 1 - Baseline: >75% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 1 - Week 52: Absent: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Right Lung Zone 1 - Week 52: Absent | 3 | 2 | 3 | 0
  Pure Ground-Glass Opacity Right Lung Zone 1 - Week 52: 1-25%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Right Lung Zone 1 - Week 52: 1-25% | 1 | 0 | 0 | 3
  Pure Ground-Glass Opacity Right Lung Zone 1 - Week 52: 26-50%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Right Lung Zone 1 - Week 52: 26-50% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 1 - Week 52: 51-75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Right Lung Zone 1 - Week 52: 51-75% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 1 - Week 52: >75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Right Lung Zone 1 - Week 52: >75% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 2 - Baseline: Absent | 3 | 2 | 4 | 1
  Pure Ground-Glass Opacity Right Lung Zone 2 - Baseline: 1-25% | 1 | 0 | 1 | 2
  Pure Ground-Glass Opacity Right Lung Zone 2 - Baseline: 26-50% | 0 | 0 | 1 | 0
  Pure Ground-Glass Opacity Right Lung Zone 2 - Baseline: 51-75% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 2 - Baseline: >75% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 2 - Week 52: Absent: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Right Lung Zone 2 - Week 52: Absent | 1 | 1 | 2 | 1
  Pure Ground-Glass Opacity Right Lung Zone 2 - Week 52: 1-25%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Right Lung Zone 2 - Week 52: 1-25% | 3 | 1 | 1 | 2
  Pure Ground-Glass Opacity Right Lung Zone 2 - Week 52: 26-50%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Right Lung Zone 2 - Week 52: 26-50% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 2 - Week 52: 51-75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Right Lung Zone 2 - Week 52: 51-75% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 2 - Week 52: >75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Right Lung Zone 2 - Week 52: >75% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 3 - Baseline: Absent | 2 | 1 | 3 | 0
  Pure Ground-Glass Opacity Right Lung Zone 3 - Baseline: 1-25% | 1 | 1 | 2 | 3
  Pure Ground-Glass Opacity Right Lung Zone 3 - Baseline: 26-50% | 1 | 0 | 1 | 0
  Pure Ground-Glass Opacity Right Lung Zone 3 - Baseline: 51-75% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 3 - Baseline: >75% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 3 - Week 52: Absent: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Right Lung Zone 3 - Week 52: Absent | 2 | 1 | 2 | 0
  Pure Ground-Glass Opacity Right Lung Zone 3 - Week 52: 1-25%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Right Lung Zone 3 - Week 52: 1-25% | 1 | 0 | 1 | 2
  Pure Ground-Glass Opacity Right Lung Zone 3 - Week 52: 26-50%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Right Lung Zone 3 - Week 52: 26-50% | 1 | 1 | 0 | 1
  Pure Ground-Glass Opacity Right Lung Zone 3 - Week 52: 51-75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Right Lung Zone 3 - Week 52: 51-75% | 0 | 0 | 0 | 0
  Pure Ground-Glass Opacity Right Lung Zone 3 - Week 52: >75%: number analyzed (Participants) | 4 | 2 | 3 | 3
  Pure Ground-Glass Opacity Right Lung Zone 3 - Week 52: >75% | 0 | 0 | 0 | 0

34. Secondary Outcome: DB Period: Pharmacokinetics: Plasma Concentration of Belumosudil and Its Metabolite (KD025m2)
Description: Plasma concentration of belumosudil and its metabolite (KD025m2) at pre-dose and 3 hours post-dose at Week 4 and 8 is reported in this outcome measure. The Lower Limit of Quantification (LLOQ) was 10 nanograms per milliliter (ng/mL).
Time Frame: Pre-dose and 3 hours post-dose at Week 4 and 8
Population: Analysis was performed on mITT population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified category. Data for this outcome measure was not planned to be collected and analyzed for placebo arm.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID
Number analyzed (Participants) | 10 | 10
ng/mL
  Belumosudil: Pre-dose at Week 4 | 162.68 (215.574) | 837.75 (874.185)
  Belumosudil: 3 hours Post-dose at Week 4: number analyzed (Participants) | 9 | 10
  Belumosudil: 3 hours Post-dose at Week 4 | 1081.56 (1093.259) | 1824.60 (1216.098)
  Belumosudil: Pre-dose at Week 8: number analyzed (Participants) | 10 | 9
  Belumosudil: Pre-dose at Week 8 | 90.74 (94.665) | 613.67 (387.507)
  Belumosudil: 3 hours Post-dose at Week 8: number analyzed (Participants) | 10 | 9
  Belumosudil: 3 hours Post-dose at Week 8 | 1367.60 (1148.820) | 1528.33 (1026.514)
  KD025m2: Pre-dose at Week 4 | 18.81 (24.451) | 71.57 (89.009)
  KD025m2: 3 hours Post-dose at Week 4: number analyzed (Participants) | 9 | 10
  KD025m2: 3 hours Post-dose at Week 4 | 131.62 (235.429) | 166.36 (175.126)
  KD025m2: Pre-dose at Week 8: number analyzed (Participants) | 10 | 9
  KD025m2: Pre-dose at Week 8 | 5.53 (9.461) | 60.47 (44.930)
  KD025m2: 3 hours Post-dose at Week 8: number analyzed (Participants) | 10 | 9
  KD025m2: 3 hours Post-dose at Week 8 | 189.23 (295.346) | 139.78 (146.559)

35. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: Adverse event (AE): any untoward medical occurrence in a participant who received study drug and did not necessarily had to have a causal relationship with the treatment. Serious adverse event (SAE) was any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs: AEs with onset after the first dose of study drug or existing AEs that worsened during TEAE Period (for DB period: From Day 1 (Week 0) up to Week 28; for OLE period: from Week 29 up to 4 weeks post last study drug administration).
Time Frame: For DB period: From Day 1 (Week 0) up to Week 28; for OLE period: from Week 29 up to 4 weeks post last study drug administration (i.e., up to Week 56)
Population: Analysis was performed on safety population which included all participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 11 | 12 | 12 | 10 | 5 | 10 | 6
Participants
  TEAEs | 11 | 11 | 11 | 9 | 5 | 9 | 5
  TESAEs | 2 | 0 | 3 | 0 | 0 | 1 | 0

36. Secondary Outcome: DB Period: Change From Baseline in Vital Signs: Systolic and Diastolic Blood Pressure at Week 24
Description: Vital signs (systolic and diastolic blood pressure) were measured with the participants after having rested in sitting position. Vital signs assessments were performed before the electrocardiogram (ECG) and other scheduled assessments. Change from Baseline in systolic and diastolic blood pressure at Week 24 was reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: Analysis was performed on safety population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure. For participants who received placebo/belumosudil in the DB period, the Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in the DB period.
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 10 | 10 | 11
millimeters of mercury
  Systolic blood pressure | 1.9 (15.13) | 3.9 (10.60) | 2.2 (8.72)
  Diastolic blood pressure | -0.9 (10.52) | 7.1 (8.95) | -0.5 (7.27)

37. Secondary Outcome: OLE: Change From Baseline in Vital Signs: Systolic and Diastolic Blood Pressure at Week 52
Description: Change from Baseline in systolic and diastolic blood pressure at Week 52 was reported in this outcome measure. Vital signs (systolic and diastolic blood pressure) were measured with the participants after having rested in sitting position. Vital signs assessments were performed before ECGs and other schedules assessments. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period.
Time Frame: Baseline, Week 52
Population: Analysis was performed on safety population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure.
Measure: Mean (Standard Deviation); unit: millimeters of mercury
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 10 | 5 | 7 | 6
millimeters of mercury
  Systolic blood pressure | -2.4 (16.30) | -1.2 (15.30) | 5.0 (16.41) | -9.5 (19.61)
  Diastolic blood pressure | -4.3 (8.06) | 0.6 (12.74) | 4.9 (9.17) | -6.2 (17.43)

38. Secondary Outcome: DB Period: Change From Baseline in Vital Signs: Pulse at Week 24
Description: Vital sign (pulse) was measured with the participants after having rested in sitting position. Vital signs assessments were performed before ECGs and other scheduled assessments. Change from Baseline in vital signs: pulse at Week 24 was reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 10 | 10 | 11
beats per minute | -3.1 (9.49) | -2.8 (13.00) | -2.0 (7.46)

39. Secondary Outcome: OLE Period: Change From Baseline in Vital Signs: Pulse at Week 52
Description: Vital sign (pulse) was measured with the participants after having rested in sitting position. Vital signs assessments were performed before ECGs and other scheduled assessments. Change from Baseline in vital signs: pulse at Week 52 was reported in this outcome measure. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period.
Time Frame: Baseline, Week 52
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 10 | 5 | 7 | 6
beats per minute | -5.9 (6.47) | -1.6 (4.39) | 1.3 (13.73) | -12.2 (34.37)

40. Secondary Outcome: DB Period: Change From Baseline in Vital Signs: Respiratory Rate at Week 24
Description: Vital sign (respiratory rate) was measured with the participants after having rested in sitting position. Vital signs assessments were performed before ECGs and other scheduled assessments. Change from Baseline in vital signs: respiratory rate at Week 24 was reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 7 | 10 | 11
breaths per minute | 1.4 (3.41) | 0.1 (2.13) | 0.6 (1.86)

41. Secondary Outcome: OLE Period: Change From Baseline in Vital Signs: Respiratory Rate at Week 52
Description: Vital sign (respiratory rate) was measured with the participants after having rested in sitting position. Vital signs assessments were performed before ECGs and other scheduled assessments. Change from Baseline in vital signs: respiratory rate at Week 52 was reported in this outcome measure. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period.
Time Frame: Baseline, Week 52
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 7 | 5 | 6 | 6
breaths per minute | 0.0 (2.31) | 1.4 (1.52) | 0.3 (1.86) | 0.0 (2.10)

42. Secondary Outcome: DB Period: Change From Baseline in 12-lead Electrocardiogram (ECG) Values: Heart Rate at Week 24
Description: ECGs were recorded after the participant had rested in the supine position for at least 5 minutes and were performed prior to any blood sample collection. Change from Baseline in 12-lead ECG values: heart rate at Week 24 was reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 10 | 10 | 11
beats per minute | -3.6 (8.71) | -2.1 (3.57) | -5.5 (10.52)

43. Secondary Outcome: OLE Period: Change From Baseline in 12-lead Electrocardiogram Values: Heart Rate at Week 52
Description: ECGs were recorded after the participant had rested in the supine position for at least 5 minutes and were performed prior to any blood sample collection. Change from Baseline in 12-lead ECG values: heart rate at Week 52 was reported in this outcome measure. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period.
Time Frame: Baseline, Week 52
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 10 | 5 | 6 | 6
beats per minute | -3.6 (10.83) | 1.0 (6.52) | -0.7 (10.88) | -13.8 (24.13)

44. Secondary Outcome: DB Period: Change From Baseline in 12-lead Electrocardiogram Values: PR Interval, RR Interval, QRS Interval, QT Interval and QTcF Interval at Week 24
Description: ECGs were recorded after the participant had rested in the supine position for at least 5 minutes and were performed prior to any blood sample collection. Change from Baseline in 12-lead ECG values: PR interval, RR interval, QRS interval, QT interval and QTcF interval at Week 24 was reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: Analysis was performed on safety population. Here, 'overall number of participants analyzed' = participants with available data for this outcome measure and 'number analyzed' = participants with available data for each specified category. For participants who received placebo/belumosudil in the DB period, the Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in the DB period.
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 10 | 10 | 11
millisecond
  PR Interval: number analyzed (Participants) | 10 | 9 | 11
  PR Interval | 2.4 (10.96) | 1.6 (9.74) | -1.4 (7.58)
  RR Interval | 46.1 (114.87) | 18.0 (39.71) | 47.2 (110.91)
  QRS Interval | 0.8 (6.55) | 0.6 (3.89) | -0.5 (8.71)
  QT Interval | 8.9 (16.87) | 7.5 (14.84) | 12.4 (23.64)
  QTcF Interval | 2.433 (12.039) | 5.008 (12.560) | 4.766 (14.177)

45. Secondary Outcome: OLE Period: Change From Baseline in 12-lead Electrocardiogram Values: PR Interval, RR Interval, QRS Interval, QT Interval and QTcF Interval at Week 52
Description: ECGs were recorded after the participant had rested in the supine position for at least 5 minutes and were performed prior to any blood sample collection. Change from Baseline in 12-lead ECG values: PR interval, RR interval, QRS interval, QT interval and QTcF interval at Week 52 was reported in this outcome measure. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period.
Time Frame: Baseline, Week 52
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: millisecond
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 10 | 5 | 6 | 6
millisecond
  PR Interval | 6.2 (8.92) | 1.6 (9.63) | 6.5 (11.66) | 7.5 (10.99)
  RR Interval | 40.3 (120.90) | -25.2 (93.73) | 18.5 (153.16) | 145.2 (251.04)
  QRS Interval | -0.2 (8.51) | 4.2 (6.83) | 0.5 (6.25) | -1.2 (4.31)
  QT Interval | 6.3 (16.76) | -0.4 (14.77) | 2.2 (22.33) | 27.5 (53.48)
  QTcF Interval | 0.056 (12.791) | 3.080 (14.850) | 0.108 (13.310) | 3.873 (17.489)

46. Secondary Outcome: DB Period: Change From Baseline in Hematological Parameters: Percentage of Basophils/Leukocytes, Eosinophils/Leukocytes, Lymphocytes/Leukocytes, Monocytes/Leukocytes and Neutrophils/Leukocytes at Week 24
Description: Blood samples were collected at specified timepoints to assess hematological parameters. Change from Baseline in hematological parameters: percentage of basophils/leukocytes, eosinophils/leukocytes, lymphocytes/leukocytes, monocytes/leukocytes and neutrophils/leukocytes at Week 24 was reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: percentage of white blood cells
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 10 | 9 | 11
percentage of white blood cells
  Basophils/Leukocytes | 0.00 (0.340) | 0.26 (0.575) | 0.04 (0.273)
  Eosinophils/Leukocytes | 0.02 (0.745) | -0.07 (1.203) | 0.50 (1.001)
  Lymphocytes/Leukocytes | -0.61 (3.618) | 3.29 (4.418) | 1.89 (7.214)
  Monocytes/Leukocytes | -0.61 (1.024) | -0.41 (2.153) | 0.22 (1.455)
  Neutrophils/Leukocytes | 1.24 (4.255) | -1.04 (8.411) | -2.60 (8.110)

47. Secondary Outcome: OLE Period: Change From Baseline in Hematological Parameters: Percentage of Basophils/Leukocytes, Eosinophils/Leukocytes, Lymphocytes/Leukocytes, Monocytes/Leukocytes and Neutrophils/Leukocytes at Week 52
Description: Blood samples were collected at specified timepoints to assess hematological parameters. Change from Baseline in hematological parameters: percentage of basophils/leukocytes, eosinophils/leukocytes, lymphocytes/leukocytes, monocytes/leukocytes and neutrophils/leukocytes at Week 52 was reported in this outcome measure. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period.
Time Frame: Baseline, Week 52
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: percentage of white blood cells
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 10 | 5 | 7 | 6
percentage of white blood cells
  Basophils/Leukocytes | 0.29 (0.341) | -0.06 (0.336) | 0.79 (0.934) | 0.00 (0.303)
  Eosinophils/Leukocytes | -0.05 (0.721) | 0.32 (0.694) | 0.36 (3.233) | 0.65 (0.737)
  Lymphocytes/Leukocytes | -1.18 (4.996) | -0.02 (6.823) | 5.80 (6.817) | 1.87 (6.490)
  Monocytes/Leukocytes | -0.22 (1.211) | -0.20 (0.797) | 0.46 (1.577) | -0.75 (2.449)
  Neutrophils/Leukocytes | 1.18 (5.401) | 0.02 (5.513) | -4.77 (7.592) | -1.75 (7.900)

48. Secondary Outcome: DB Period: Change From Baseline in Hematological Parameter: Hematocrit at Week 24
Description: Blood samples were collected at specified timepoints to assess hematological parameters. Change from Baseline in hematological parameter (hematocrit, fraction of 1.0) at Week 24 was reported in this outcome measure. The hematocrit is percentage of the volume of whole blood that is made up of red blood cells.
Time Frame: Baseline, Week 24
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: percentage of red blood cells in blood
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 10 | 9 | 11
percentage of red blood cells in blood | 0.002 (0.027) | 0.003 (0.040) | 0.012 (0.067)

49. Secondary Outcome: OLE Period: Change From Baseline in Hematological Parameter: Hematocrit at Week 52
Description: Blood samples were collected at specified timepoints to assess hematological parameters. Change from Baseline in hematological parameter (hematocrit, fraction of 1.0) at Week 52 was reported in this outcome measure. The hematocrit is percentage of the volume of whole blood that is made up of red blood cells. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period.
Time Frame: Baseline, Week 52
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: percentage of red blood cells in blood
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 10 | 5 | 7 | 6
percentage of red blood cells in blood | -0.004 (0.033) | -0.024 (0.042) | -0.003 (0.023) | -0.032 (0.026)

50. Secondary Outcome: DB Period: Change From Baseline in Hematological Parameter: Hemoglobin at Week 24
Description: Blood samples were collected at specified timepoints to assess hematological parameters. Change from Baseline in hematological parameter: hemoglobin at Week 24 was reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 10 | 9 | 11
grams per liter | 1.2 (7.39) | -3.6 (14.77) | 2.6 (19.96)

51. Secondary Outcome: OLE Period: Change From Baseline in Hematological Parameter: Hemoglobin at Week 52
Description: Blood samples were collected at specified timepoints to assess hematological parameters. Change from Baseline in hematological parameter: hemoglobin at Week 52 was reported in this outcome measure. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period.
Time Frame: Baseline, Week 52
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 10 | 5 | 7 | 6
grams per liter | -2.4 (8.45) | -2.8 (12.01) | 0.4 (6.70) | -8.0 (10.49)

52. Secondary Outcome: DB Period: Change From Baseline in Hematological Parameter: Erythrocytes Mean Corpuscular Volume at Week 24
Description: Blood samples were collected at specified timepoints to assess hematological parameters. Change from Baseline in hematological parameter: erythrocytes mean corpuscular volume at Week 24 was reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: femtoliters
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 10 | 9 | 11
femtoliters | -0.7 (2.00) | 2.2 (3.15) | 0.5 (2.70)

53. Secondary Outcome: OLE Period: Change From Baseline in Hematological Parameter: Erythrocytes Mean Corpuscular Volume at Week 52
Description: Blood samples were collected at specified timepoints to assess hematological parameters. Change from Baseline in hematological parameter: erythrocytes mean corpuscular volume at Week 52 was reported in this outcome measure. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period.
Time Frame: Baseline, Week 52
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: femtoliters
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 10 | 5 | 7 | 6
femtoliters | -0.2 (2.20) | -0.6 (1.34) | 0.7 (2.56) | -3.3 (4.03)

54. Secondary Outcome: DB Period: Change From Baseline in Hematological Parameter: Platelets at Week 24
Description: Blood samples were collected at specified timepoints to assess hematological parameters. Change from Baseline in hematological parameter: platelets at Week 24 was reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 10 | 9 | 11
10^9 cells per liter | -2.8 (69.88) | -29.3 (56.97) | -28.1 (64.79)

55. Secondary Outcome: OLE Period: Change From Baseline in Hematological Parameter: Platelets at Week 52
Description: Blood samples were collected at specified timepoints to assess hematological parameters. Change from Baseline in hematological parameter: platelets at Week 52 was reported in this outcome measure. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period.
Time Frame: Baseline, Week 52
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 10 | 5 | 7 | 6
10^9 cells per liter | -5.9 (59.12) | -25.6 (65.23) | -31.3 (62.38) | 60.7 (95.98)

56. Secondary Outcome: DB Period: Change From Baseline in Hematological Parameter: Erythrocytes at Week 24
Description: Blood samples were collected at specified timepoints to assess hematological parameters. Change from Baseline in hematological parameter: erythrocytes at Week 24 was reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 10 | 9 | 11
10^12 cells per liter | 0.05 (0.331) | -0.07 (0.480) | 0.12 (0.666)

57. Secondary Outcome: OLE Period: Change From Baseline in Hematological Parameter: Erythrocytes at Week 52
Description: Blood samples were collected at specified timepoints to assess hematological parameters. Change from Baseline in hematological parameter: erythrocytes at Week 52 was reported in this outcome measure. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period.
Time Frame: Baseline, Week 52
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: 10^12 cells per liter
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 10 | 5 | 7 | 6
10^12 cells per liter | -0.06 (0.337) | -0.18 (0.409) | -0.09 (0.227) | -0.17 (0.163)

58. Secondary Outcome: DB Period: Change From Baseline in Hematological Parameter: Leukocytes at Week 24
Description: Blood samples were collected at specified timepoints to assess hematological parameters. Change from Baseline in hematological parameter: leukocytes at Week 24 was reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 10 | 9 | 11
10^9 cells per liter | -0.579 (1.030) | -0.673 (2.427) | -0.124 (1.310)

59. Secondary Outcome: OLE Period: Change From Baseline in Hematological Parameter: Leukocytes at Week 52
Description: Blood samples were collected at specified timepoints to assess hematological parameters. Change from Baseline in hematological parameter: leukocytes at Week 52 was reported in this outcome measure. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period.
Time Frame: Baseline, Week 52
Population: as for outcome 37
Measure: Mean (Standard Deviation); unit: 10^9 cells per liter
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 10 | 5 | 7 | 6
10^9 cells per liter | -0.255 (1.519) | -0.386 (0.198) | -2.281 (4.379) | -1.015 (1.382)

60. Secondary Outcome: DB Period: Change From Baseline in Clinical Chemistry Parameter: Albumin, Globulin and Protein at Week 24
Description: Blood samples were collected at specified timepoints to assess clinical chemistry parameters. Change from Baseline in clinical chemistry parameter: albumin, globulin and protein at Week 24 was reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: Analysis was performed on safety population. Here, 'overall number of participants analyzed' = participants with available data. For participants who received placebo/belumosudil in the DB period, the Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in the DB period.
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 10 | 10 | 11
grams per liter
  Albumin | -0.3 (1.83) | 0.1 (2.42) | -0.9 (2.39)
  Globulin | -1.5 (1.43) | 0.0 (2.71) | -2.7 (10.20)
  Protein | -1.8 (3.05) | 0.1 (3.75) | -3.6 (9.07)

61. Secondary Outcome: OLE Period: Change From Baseline in Clinical Chemistry Parameter: Albumin, Globulin and Protein at Week 52
Description: Blood samples were collected at specified timepoints to assess clinical chemistry parameters. Change from Baseline in clinical chemistry parameter: albumin, globulin and protein at Week 52 was reported in this outcome measure. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period.
Time Frame: Baseline, Week 52
Population: Analysis was performed on safety population. Here, 'overall number of participants analyzed' = participants with available data.
Measure: Mean (Standard Deviation); unit: grams per liter
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 9 | 5 | 7 | 6
grams per liter
  Albumin | -1.3 (3.20) | -1.0 (2.65) | 0.0 (3.06) | -0.8 (2.14)
  Globulin | -3.4 (2.83) | -0.8 (1.92) | 0.0 (2.83) | 0.5 (5.68)
  Protein | -4.8 (4.68) | -1.8 (2.49) | 0.0 (4.90) | -0.3 (4.50)

62. Secondary Outcome: DB Period: Change From Baseline in Clinical Chemistry Parameter: Alkaline Phosphatase, Alanine Aminotransferase, Aspartate Aminotransferase, Creatine Kinase, Gamma Glutamyl Transferase, and Lactate Dehydrogenase at Week 24
Description: Blood samples were collected at specified timepoints to assess clinical chemistry parameters. Change from Baseline in clinical chemistry parameter: alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, creatine kinase, gamma-glutamyl transferase, and lactate dehydrogenase at Week 24 was reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: Analysis was performed on safety population. Here, 'overall number of participants analyzed' = participants with available data and 'number analyzed' = participants with available data for each specified category. For participants who received placebo/belumosudil in the DB period, the Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in the DB period.
Measure: Mean (Standard Deviation); unit: units per liter
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 10 | 10 | 11
units per liter
  Alkaline Phosphatase | -1.7 (14.46) | 1.3 (7.76) | 4.1 (9.31)
  Alanine Aminotransferase: number analyzed (Participants) | 10 | 9 | 11
  Alanine Aminotransferase | 1.9 (7.87) | -6.9 (16.84) | 0.4 (13.51)
  Aspartate Aminotransferase: number analyzed (Participants) | 10 | 9 | 11
  Aspartate Aminotransferase | 0.6 (5.17) | -6.9 (18.18) | 0.1 (7.48)
  Creatine Kinase: number analyzed (Participants) | 10 | 9 | 11
  Creatine Kinase | 16.9 (124.46) | -15.6 (83.11) | -1.7 (29.99)
  Gamma Glutamyl Transferase | 0.1 (7.67) | -0.8 (8.72) | 1.1 (6.99)
  Lactate Dehydrogenase: number analyzed (Participants) | 8 | 7 | 9
  Lactate Dehydrogenase | 6.9 (33.88) | -19.0 (28.33) | 6.7 (14.52)

63. Secondary Outcome: OLE Period: Change From Baseline in Clinical Chemistry Parameter: Alkaline Phosphatase, Alanine Aminotransferase, Aspartate Aminotransferase, Creatine Kinase, Gamma Glutamyl Transferase, and Lactate Dehydrogenase at Week 52
Description: Blood samples were collected at specified timepoints to assess clinical chemistry parameters. Change from Baseline in clinical chemistry parameter: alkaline phosphatase, alanine aminotransferase, aspartate aminotransferase, creatine kinase, gamma-glutamyl transferase, and lactate dehydrogenase at Week 52 was reported in this outcome measure. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period.
Time Frame: Baseline, Week 52
Population: Analysis was performed on safety population. Here, 'overall number of participants analyzed' = participants with available data and 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: units per liter
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 9 | 5 | 7 | 6
units per liter
  Alkaline Phosphatase | 0.9 (18.00) | -4.2 (9.23) | 2.3 (12.57) | 7.5 (17.06)
  Alanine Aminotransferase | 5.0 (11.93) | 2.2 (2.17) | -5.0 (18.41) | 1.2 (5.04)
  Aspartate Aminotransferase | 3.2 (9.83) | 0.4 (2.30) | -3.9 (22.41) | -3.5 (3.51)
  Creatine Kinase | 10.0 (79.24) | 26.6 (42.34) | 16.7 (92.29) | -16.2 (20.01)
  Gamma Glutamyl Transferase | 0.7 (5.61) | -0.8 (1.30) | -6.1 (14.09) | -1.2 (9.97)
  Lactate Dehydrogenase: number analyzed (Participants) | 8 | 5 | 6 | 6
  Lactate Dehydrogenase | 4.3 (51.53) | -8.8 (20.66) | -13.5 (37.95) | -39.8 (73.03)

64. Secondary Outcome: DB Period: Change From Baseline in Clinical Chemistry Parameter: Bicarbonate, Blood Urea Nitrogen, Calcium, Chloride, Glucose, Potassium, Magnesium, Phosphate and Sodium at Week 24
Description: Blood samples were collected at specified timepoints to assess clinical chemistry parameters. Change from Baseline in clinical chemistry parameter: bicarbonate, blood urea nitrogen, calcium, chloride, glucose, potassium, magnesium, phosphate and sodium at Week 24 was reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: millimoles per liter
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 10 | 10 | 11
millimoles per liter
  Bicarbonate | -1.83 (2.058) | 0.42 (0.935) | 0.48 (1.946)
  Blood Urea Nitrogen | -0.011 (0.163) | -0.086 (0.224) | 0.005 (0.163)
  Calcium | -0.022 (0.102) | 0.005 (0.068) | -0.033 (0.059)
  Chloride | -0.4 (2.32) | -0.3 (1.64) | 1.2 (1.40)
  Glucose | -0.304 (1.260) | -0.767 (1.236) | -0.219 (1.016)
  Potassium: number analyzed (Participants) | 10 | 9 | 11
  Potassium | -0.11 (0.555) | 0.04 (0.388) | -0.04 (0.229)
  Magnesium | -0.005 (0.071) | -0.011 (0.055) | 0.000 (0.053)
  Phosphate | -0.113 (0.167) | 0.076 (0.093) | -0.085 (0.127)
  Sodium | -1.4 (2.01) | 0.7 (1.57) | 0.5 (1.44)

65. Secondary Outcome: OLE Period: Change From Baseline in Clinical Chemistry Parameter: Bicarbonate, Blood Urea Nitrogen, Calcium, Chloride, Glucose, Potassium, Magnesium, Phosphate and Sodium at Week 52
Description: Blood samples were collected at specified timepoints to assess clinical chemistry parameters. Change from Baseline in clinical chemistry parameter: bicarbonate, blood urea nitrogen, calcium, chloride, glucose, potassium, magnesium, phosphate and sodium at Week 52 was reported in this outcome measure. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period.
Time Frame: Baseline, Week 52
Population: as for outcome 61
Measure: Mean (Standard Deviation); unit: millimoles per liter
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 9 | 5 | 7 | 6
millimoles per liter
  Bicarbonate | -1.60 (1.572) | 1.90 (1.414) | 0.63 (3.256) | 0.53 (1.998)
  Blood Urea Nitrogen | -0.008 (0.127) | 0.094 (0.206) | -0.026 (0.130) | -0.030 (0.139)
  Calcium | -0.074 (0.082) | -0.010 (0.065) | -0.006 (0.128) | -0.027 (0.080)
  Chloride | 0.4 (1.81) | -1.4 (2.07) | 1.4 (2.88) | -0.7 (1.03)
  Glucose | -0.147 (1.080) | 0.612 (1.063) | -0.319 (0.700) | 0.092 (1.330)
  Potassium | -0.18 (0.441) | 0.00 (0.469) | 0.01 (0.518) | -0.23 (0.273)
  Magnesium | -0.028 (0.079) | -0.058 (0.025) | -0.013 (0.045) | -0.007 (0.030)
  Phosphate | -0.108 (0.137) | 0.016 (0.116) | 0.124 (0.126) | 0.037 (0.086)
  Sodium | -1.1 (2.62) | 0.2 (0.45) | 1.3 (2.56) | -1.3 (1.03)

66. Secondary Outcome: DB Period: Change From Baseline in Clinical Chemistry Parameter: Direct Bilirubin, Bilirubin, Creatinine and Urate at Week 24
Description: Blood samples were collected at specified timepoints to assess clinical chemistry parameters. Change from Baseline in clinical chemistry parameter: direct bilirubin, bilirubin, creatinine and urate at Week 24 was reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: as for outcome 62
Measure: Mean (Standard Deviation); unit: micromole per liter
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 10 | 10 | 11
micromole per liter
  Direct Bilirubin: number analyzed (Participants) | 10 | 8 | 11
  Direct Bilirubin | 0.171 (0.541) | -0.214 (0.996) | -0.233 (0.553)
  Bilirubin | 1.026 (2.308) | 1.368 (2.251) | -0.466 (2.767)
  Creatinine | 3.536 (7.455) | 2.652 (14.466) | -3.215 (9.078)
  Urate | -4.760 (44.860) | -6.545 (31.164) | 4.868 (43.383)

67. Secondary Outcome: OLE Period: Change From Baseline in Clinical Chemistry Parameter: Direct Bilirubin, Bilirubin, Creatinine and Urate at Week 52
Description: Blood samples were collected at specified timepoints to assess clinical chemistry parameters. Change from Baseline in clinical chemistry parameter: direct bilirubin, bilirubin, creatinine and urate at Week 52 was reported in this outcome measure. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period.
Time Frame: Baseline, Week 52
Population: as for outcome 61
Measure: Mean (Standard Deviation); unit: micromole per liter
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 9 | 5 | 7 | 6
micromole per liter
  Direct Bilirubin | 0.285 (0.605) | -0.171 (0.382) | -0.489 (0.969) | -0.428 (1.047)
  Bilirubin | 0.950 (2.280) | -1.026 (0.937) | 0.489 (2.144) | 0.285 (2.517)
  Creatinine | 8.840 (9.883) | 8.840 (6.251) | 2.526 (9.836) | 0.000 (5.591)
  Urate | 2.644 (41.768) | 2.380 (14.934) | 6.800 (45.109) | -15.867 (47.102)

68. Secondary Outcome: DB Period: Change From Baseline in Clinical Chemistry Parameter: Calcium Corrected at Week 24
Description: Blood samples were collected at specified timepoints to assess clinical chemistry parameters. Change from Baseline in clinical chemistry parameter: calcium corrected at Week 24 was reported in this outcome measure.
Time Frame: Baseline, Week 24
Population: as for outcome 60
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 10 | 10 | 11
milligrams per deciliter | -0.06 (0.303) | 0.00 (0.249) | -0.05 (0.211)

69. Secondary Outcome: OLE Period: Change From Baseline in Clinical Chemistry Parameter: Calcium Corrected at Week 52
Description: Blood samples were collected at specified timepoints to assess clinical chemistry parameters. Change from Baseline in clinical chemistry parameter: calcium corrected at Week 52 was reported in this outcome measure. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period.
Time Frame: Baseline, Week 52
Population: as for outcome 61
Measure: Mean (Standard Deviation); unit: milligrams per deciliter
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 9 | 5 | 7 | 6
milligrams per deciliter | -0.18 (0.222) | 0.08 (0.192) | -0.03 (0.454) | -0.05 (0.373)

70. Secondary Outcome: DB Period: Change From Baseline in Clinical Chemistry Parameter: Glomerular Filtration Rate at Week 24
Description: Blood samples were collected at specified timepoints to assess clinical chemistry parameters. Change from Baseline in clinical chemistry parameter: glomerular filtration rate at Week 24 was reported in this outcome measure. Expanded unit of measure is milliliter per minute per 1.73 square meters.
Time Frame: Baseline, Week 24
Population: as for outcome 60
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo
Number analyzed (Participants) | 5 | 5 | 7
mL/min/1.73 m^2 | -4.76 (11.414) | -6.88 (11.749) | 3.36 (10.229)

71. Secondary Outcome: OLE Period: Change From Baseline in Clinical Chemistry Parameter: Glomerular Filtration Rate at Week 52
Description: Blood samples were collected at specified timepoints to assess clinical chemistry parameters. Change from Baseline in clinical chemistry parameter: glomerular filtration rate at Week 52 was reported in this outcome measure. Participants who received placebo in DB period and re-randomized into OLE period, OLE period Baseline was defined as valid and last non-missing value obtained prior to participant receiving first dose of belumosudil in OLE period. Participants who received belumosudil in DB period and continued belumosudil in OLE period, Baseline value was defined as valid and last non-missing value obtained within 29 days prior to participant receiving first study medication in DB period.
Time Frame: Baseline, Week 52
Population: as for outcome 61
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
Number analyzed (Participants) | 1 | 1 | 1 | 2
mL/min/1.73 m^2 | -26.60 | -16.40 | -0.40 | -9.70 (13.152)

ADVERSE EVENTS:
Time Frame: For DB period: From Day 1 (Week 0) up to Week 28; for OLE period: from Week 29 up to 4 weeks post last study drug administration (i.e., up to Week 56)
Description: Analysis was performed on safety population.
Arm/Group | DB Period: Belumosudil QD | DB Period: Belumosudil BID | DB Period: Placebo | OLE Period: Belumosudil QD | OLE Period: Placebo/Belumosudil QD | OLE Period: Belumosudil BID | OLE Period: Placebo/Belumosudil BID
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12 | 0/12 | 0/10 | 0/5 | 0/10 | 0/6
Serious Adverse Events (participants affected / at risk) | 2/11 | 0/12 | 3/12 | 0/10 | 0/5 | 1/10 | 0/6
Other Adverse Events (participants affected / at risk) | 10/11 | 11/12 | 11/12 | 9/10 | 5/5 | 9/10 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB Period: Belumosudil QD (N=11) | DB Period: Belumosudil BID (N=12) | DB Period: Placebo (N=12) | OLE Period: Belumosudil QD (N=10) | OLE Period: Placebo/Belumosudil QD (N=5) | OLE Period: Belumosudil BID (N=10) | OLE Period: Placebo/Belumosudil BID (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial Flutter (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac Failure Congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scleroderma Renal Crisis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DB Period: Belumosudil QD (N=11) | DB Period: Belumosudil BID (N=12) | DB Period: Placebo (N=12) | OLE Period: Belumosudil QD (N=10) | OLE Period: Placebo/Belumosudil QD (N=5) | OLE Period: Belumosudil BID (N=10) | OLE Period: Placebo/Belumosudil BID (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mastocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bundle Branch Block Right (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Supraventricular Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival Haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye Inflammation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision Blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 1 (1) | 2 (2) | 1 (1) | 2 (3) | 1 (1) | 1 (3)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Angiodysplasia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (8) | 0 (0) | 5 (5) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (5) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Calcinosis (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Early Satiety (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Influenza Like Illness (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema Peripheral (General disorders) | 1 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Peripheral Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sensation Of Foreign Body (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder Disorder (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Covid-19 (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis Streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-Acute Covid-19 Syndrome (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory Tract Infection Viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental Restoration Failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iliotibial Band Syndrome (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Traumatic Ulcer (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood Creatine Phosphokinase Increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Pressure Increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram Qt Prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram Abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sars-Cov-2 Test Positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin C Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin D Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Increased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin B12 Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendon Disorder (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0)
Tenosynovitis Stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasal Neoplasm Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carpal Tunnel Syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 2 (3) | 0 (0) | 7 (11) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory Impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Trigeminal Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Breast Mass (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Macule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Precancerous Skin Lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Hypertrophy (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Raynaud's Phenomenon (Vascular disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated early by the Sponsor due to slow enrollment and strategic consideration and was not driven due to any safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-05-27): https://cdn.clinicaltrials.gov/large-docs/99/NCT03919799/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-29): https://cdn.clinicaltrials.gov/large-docs/99/NCT03919799/SAP_001.pdf